CLINICAL TRIAL: NCT00976820
Title: A Study to Evaluate the Safety and Immunogenicity of A/California/7/2009 (H1N1)V-like Vaccines GSK2340274A and GSK2340273A in Children 6 Months to Less Than 9 Years of Age
Brief Title: Safety and Immunogenicity of H1N1 Vaccines in Children Aged 6 Months to Less Than 9 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113482
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-07

CONDITIONS: Influenza
Keywords: influenza infection; Influenza Vaccines; GSK Bio's influenza vaccine GSK2340273A; GSK Bio's influenza vaccine GSK2340274A
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Arepanrix/F1 Group (Experimental): Subjects, aged 6 months - 9 years, male or female, received 2 doses of Arepanrix™-formulation 1 (F1) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh [for children under (<) 12 months of age]. The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
  Interventions: Biological: GSK2340274A
- Arepanrix/F2 Group (Experimental): Subjects, aged 6 months - 9 years, male or female, received 2 doses of Arepanrix™-formulation 2 (F2) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
  Interventions: Biological: GSK2340274A
- GSK2340273A/F1 Group (Experimental): Subjects, aged 6 months - 9 years, male or female, received 2 doses of GSK2340273A-formulation 1 (F1) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
  Interventions: Biological: GSK2340273A
- GSK2340273A/F2 Group (Experimental): Subjects, aged 6 months - 9 years, male or female, received 2 doses of GSK2340273A-formulation 2 (F2) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
  Interventions: Biological: GSK2340273A

INTERVENTIONS:
Biological: GSK2340274A — Two intramuscular injections
  Arms: Arepanrix/F1 Group; Arepanrix/F2 Group
Biological: GSK2340273A — Two intramuscular injections
  Arms: GSK2340273A/F1 Group; GSK2340273A/F2 Group

SUMMARY:
The purpose of this study is to characterize the safety and immune response of the H1N1 (swine) flu vaccines GSK2340274A and GSK2340273A in children 6 months to less than 9 years of age.

This Protocol Posting has been updated following the Protocol amendment 1 & 2, September and October 2009. The sections impacted are study design, objectives and analysis methods.

DETAILED DESCRIPTION:
Collaborators: United States Department of Health and Human Services, Office of Biomedical Advanced Research and Development Authority

ELIGIBILITY:
Inclusion Criteria:

* Male or female children 6 months to less than 9 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject's parent/ legally acceptable representative (LAR); written informed assent obtained from the subject if appropriate.
* Good general health as established by medical history and clinical examination before entering into the study.
* Safety laboratory test results within the parameters specified in the protocol.
* Parent/ LAR access to a consistent means of telephone contact, land line or mobile, but NOT a pay phone or other multiple-user device.
* Subjects who the investigator believes that their parent(s)/ LAR can and will comply with the requirements of the protocol.
* Female subjects of non-childbearing potential (pre-menarche) may be enrolled in the study.

Exclusion Criteria:

* Previous vaccination with an H1N1v-like virus vaccine or a medical history of physician-confirmed infection with an H1N1v-like virus.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, even if stable, are deemed by the investigator to render the potential subject or parent(s)/ LAR(s) unable/unlikely to provide accurate safety reports.
* Presence of a temperature >= 38.0ºC (>=100.4ºF) by any route or method, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Receipt of systemic glucocorticoids within 1 month prior to study enrollment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment. Topical, intra-articular or inhaled glucocorticoids are allowed.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrollment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin are eligible if no such doses are given in the 24 hours before a study vaccination. Persons receiving prophylactic antiplatelet medications, e.g., low-dose acetylsalicylic acid, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome within 6 weeks of receipt of seasonal influenza vaccine.
* Administration of any licensed vaccine within 4 weeks before the first dose of study vaccine, with the exception of seasonal influenza vaccine.
* Planned administration of any vaccine not foreseen by the study protocol between Day 0 and the Day 42 phlebotomy, including seasonal influenza vaccine. Routine childhood vaccinations are exempted if they cannot be delayed, but they must not be administered on the same day as the H1N1 vaccine candidate.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Child in care.

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 323 (Actual)
Dates: Start 2009-10-20 (Actual); Primary Completion 2011-03-21 (Actual); Study Completion 2011-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (29):
- United States (17):
  - GSK Investigational Site, Conway, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Angelo, Texas
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, South Jordan, Utah
- Canada (12):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Langley JM, Reich D, Aggarwal N, Connor D, Lebel MH, Gupta A, Garfield H, Li P, Madan A, Vaughn DW. Randomized, multicenter trial of a single dose of AS03-adjuvanted or unadjuvanted H1N1 2009 pandemic influenza vaccine in children 6 months to <9 years of age: safety and immunogenicity. Pediatr Infect Dis J. 2012 Aug;31(8):848-58. doi: 10.1097/INF.0b013e31825e6cd6. PMID 22801094
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113482 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113482 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113482 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113482 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113482 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113482 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 323 subjects originally enrolled in the study, 1 subject was not included in the Total Vaccinated Cohort.
Period: Overall Study
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Started | 67 | 128 | 64 | 63
Completed | 59 | 108 | 60 | 56
Not Completed | 8 | 20 | 4 | 7
Not completed — Lost to Follow-up | 5 | 16 | 2 | 3
Not completed — Poor Compliance. Numerous Visits Booked | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Arepanrix/F1 Group: Subjects, aged 6 months - 9 years, male or female, received 2 doses of Arepanrix™-formulation 1 (F1) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- Total: Total of all reporting groups
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group | Total
Number analyzed (Participants) | 67 | 128 | 64 | 63 | 322
Age, Continuous [Mean (Standard Deviation); unit: Months] | 53.6 (31.6) | 47.4 (28.6) | 50.3 (29.0) | 54.4 (30.4) | 50.6 (29.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 58 | 33 | 30 | 148
  Male | 40 | 70 | 31 | 33 | 174
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 1 | 7 | 1 | 1 | 10
  American Indian or Alaskan native | 1 | 6 | 1 | 2 | 10
  Asian - Central/South Asian heritage | 14 | 16 | 16 | 14 | 60
  Asian - East Asian heritage | 2 | 4 | 0 | 2 | 8
  Asian - South East Asian heritage | 3 | 1 | 2 | 2 | 8
  White - Arabic/North African heritage | 0 | 3 | 0 | 1 | 4
  White - Caucasian/European heritage | 46 | 86 | 44 | 38 | 214
  Not specified | 0 | 5 | 0 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects Against Flu A/CAL/7/09 Influenza Strain - Preliminary Analysis
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination reciprocal hemagglutination inhibition (HI) titer lower than (<) 10 and a post-vaccination reciprocal HI titer higher than or equal to (≥) 40, or a pre-vaccination reciprocal hemagglutination inhibition (HI) titer ≥ 10 and at least a 4-fold increase in post vaccination reciprocal titer against the vaccine virus.
Time Frame: At Day 21
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects who received at least 1 study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 63 | 55 | 58 | 60
Participants | 60 | 53 | 45 | 36

2. Primary Outcome: Number of Seroconverted Subjects Against Flu A/CAL/7/09 Influenza Strain - First Analysis
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination reciprocal HI titer < 10 and a post-vaccination reciprocal titer higher than or equal to (≥) 40, or a pre-vaccination reciprocal hemagglutination inhibition (HI) titer ≥ 10 and at least a 4-fold increase in post vaccination reciprocal titer against the vaccine virus.
Time Frame: At Day 21
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity at Day 21, which included all evaluable subjects who met all eligibility criteria, who complied with the protocol requirements and for whom immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 57 | 47 | 55 | 57
Participants | 54 | 45 | 41 | 34

3. Primary Outcome: Number of Seroconverted Subjects Against Flu A/CAL/7/09 Influenza Strain - Second Analysis
Description: as for outcome 2
Time Frame: At Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 59 | 101 | 54 | 57
Participants | 56 | 98 | 41 | 34

4. Primary Outcome: Number of Seroconverted Subjects Against Flu A/CAL/7/09 Influenza Strain - First Analysis
Description: as for outcome 2
Time Frame: At Day 42
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity at Day 42, which included all evaluable subjects who met all eligibility criteria, who complied with the protocol requirements and for whom immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 43 | 40 | 46 | 44
Participants | 43 | 39 | 46 | 38

5. Primary Outcome: Number of Seroconverted Subjects Against Flu A/CAL/7/09 Influenza Strain - Second Analysis
Description: as for outcome 2
Time Frame: At Day 42
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 44 | 84 | 46 | 44
Participants | 44 | 83 | 46 | 38

6. Primary Outcome: Number of Seroprotected Subjects Against Flu A/CAL/7/09 Influenza Strain - Preliminary Analysis
Description: A seroprotected subject was defined as a vaccinated subject with reciprocal HI titers higher than or equal to (≥) 40 against the tested virus.
Time Frame: At Day 0
Population: The analysis was performed on the Total Vaccinated Cohort at Day 21, which included all subjects who received at least 1 study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 66 | 59 | 61 | 62
Participants | 13 | 3 | 12 | 15

7. Primary Outcome: Number of Seroprotected Subjects Against Flu A/CAL/7/09 Influenza Strain - Preliminary Analysis
Description: as for outcome 6
Time Frame: At Day 21
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 63 | 56 | 59 | 60
Participants | 62 | 55 | 46 | 39

8. Primary Outcome: Number of Seroprotected Subjects Against Flu A/CAL/7/09 Influenza Strain - First Analysis
Description: as for outcome 6
Time Frame: At Day 0
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 57 | 49 | 55 | 58
Participants | 12 | 2 | 12 | 14

9. Primary Outcome: Number of Seroprotected Subjects Against Flu A/CAL/7/09 Influenza Strain - First Analysis
Description: as for outcome 6
Time Frame: At Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 57 | 49 | 55 | 57
Participants | 56 | 48 | 42 | 37

10. Primary Outcome: Number of Seroprotected Subjects Against Flu A/CAL/7/09 Influenza Strain - Second Analysis
Description: as for outcome 6
Time Frame: At Day 0
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 59 | 102 | 54 | 58
Participants | 12 | 24 | 12 | 14

11. Primary Outcome: Number of Seroprotected Subjects Against Flu A/CAL/7/09 Influenza Strain - Second Analysis
Description: as for outcome 6
Time Frame: At Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 59 | 103 | 54 | 57
Participants | 58 | 102 | 42 | 37

12. Primary Outcome: Number of Seroprotected Subjects Against Flu A/CAL/7/09 Strain - First Analysis
Description: as for outcome 6
Time Frame: At Day 0
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 43 | 40 | 46 | 44
Participants | 8 | 1 | 9 | 9

13. Primary Outcome: Number of Seroprotected Subjects Against Flu A/CAL/7/09 Influenza Strain - First Analysis
Description: as for outcome 6
Time Frame: At Day 42
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 43 | 42 | 46 | 44
Participants | 43 | 42 | 46 | 41

14. Primary Outcome: Number of Seroprotected Subjects Against Flu A/CAL/7/09 Strain - Second Analysis
Description: as for outcome 6
Time Frame: At Day 0
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 44 | 84 | 46 | 44
Participants | 8 | 20 | 9 | 9

15. Primary Outcome: Number of Seroprotected Subjects Against Flu A/CAL/7/09 Influenza Strain - Second Analysis
Description: as for outcome 6
Time Frame: At Day 42
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 44 | 87 | 46 | 44
Participants | 44 | 87 | 46 | 41

16. Primary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/CAL/7/09 Influenza Strain - Preliminary Analysis
Description: SCF was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer for the vaccine virus.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 63 | 55 | 58 | 60
Fold change | 38.6 [28.8 to 51.8] | 39.2 [29.2 to 52.5] | 14.4 [10.2 to 20.4] | 7.8 [5.6 to 11.0]

17. Primary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/CAL/7/09 Influenza Strain - First Analysis
Description: as for outcome 16
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 57 | 47 | 55 | 57
Fold change | 35.9 [26.4 to 49.0] | 40.8 [29.7 to 56.2] | 13.2 [9.2 to 18.8] | 7.6 [5.4 to 10.6]

18. Primary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/CAL/7/09 Influenza Strain - Second Analysis
Description: as for outcome 16
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 59 | 101 | 54 | 57
Fold change | 36.2 [26.8 to 48.9] | 33.6 [27.3 to 41.3] | 13.8 [9.7 to 19.6] | 7.6 [5.4 to 10.6]

19. Primary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/CAL/7/09 Influenza Strain - First Analysis
Description: as for outcome 16
Time Frame: At Day 42
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 43 | 40 | 46 | 44
Fold change | 155.3 [105.7 to 228.2] | 217.2 [163.9 to 287.9] | 44.2 [30.6 to 63.9] | 24.1 [15.9 to 36.5]

20. Primary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/CAL/7/09 Influenza Strain - Second Analysis
Description: as for outcome 16
Time Frame: At Day 42
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 44 | 84 | 46 | 44
Fold change | 157.1 [107.8 to 228.9] | 151.6 [114.0 to 201.6] | 44.2 [30.6 to 63.9] | 24.1 [15.9 to 36.5]

21. Secondary Outcome: Number of Seropositive Subjects for HI Antibodies - Preliminary Analysis
Description: A seropositive subject was defined as a subject with antibody titers greater than or equal to (≥) 1:10. The vaccine strain assessed was Flu A/CAL/7/09.
Time Frame: At Day 0 (PRE) and at Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 66 | 59 | 61 | 62
Participants
  Flu A/CAL/7/09, PRE | 17 | 4 | 13 | 15
  Flu A/CAL/7/09, D21: number analyzed (Participants) | 63 | 56 | 59 | 60
  Flu A/CAL/7/09, D21 | 63 | 56 | 57 | 56

22. Secondary Outcome: Number of Seropositive Subjects for HI Antibodies - First Analysis
Description: as for outcome 21
Time Frame: At Day 0 (PRE) and at Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 57 | 49 | 55 | 58
Participants
  Flu A/CAL/7/09, PRE | 15 | 3 | 13 | 14
  Flu A/CAL/7/09, D21: number analyzed (Participants) | 57 | 49 | 55 | 57
  Flu A/CAL/7/09, D21 | 57 | 49 | 53 | 54

23. Secondary Outcome: Number of Seropositive Subjects for HI Antibodies - Second Analysis
Description: as for outcome 21
Time Frame: At Day 0 (PRE) and at Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 59 | 103 | 54 | 58
Participants
  Flu A/CAL/7/09, PRE: number analyzed (Participants) | 59 | 102 | 54 | 58
  Flu A/CAL/7/09, PRE | 15 | 27 | 13 | 14
  Flu A/CAL/7/09, D21: number analyzed (Participants) | 59 | 103 | 54 | 57
  Flu A/CAL/7/09, D21 | 59 | 103 | 53 | 54

24. Secondary Outcome: Number of Seropositive Subjects for HI Antibodies - First Analysis
Description: as for outcome 21
Time Frame: At Day 0 (PRE) and at Day 42
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 43 | 42 | 46 | 44
Participants
  Flu A/CAL/7/09, PRE: number analyzed (Participants) | 43 | 40 | 46 | 44
  Flu A/CAL/7/09, PRE | 10 | 2 | 10 | 9
  Flu A/CAL/7/09, D42 | 43 | 42 | 46 | 44

25. Secondary Outcome: Number of Seropositive Subjects for HI Antibodies - Second Analysis
Description: as for outcome 21
Time Frame: At Day 0 (PRE) and at Day 42
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 44 | 87 | 46 | 44
Participants
  Flu A/CAL/7/09, PRE: number analyzed (Participants) | 44 | 84 | 46 | 44
  Flu A/CAL/7/09, PRE | 10 | 23 | 10 | 9
  Flu A/CAL/7/09, D42 | 44 | 87 | 46 | 44

26. Secondary Outcome: Number of Seropositive Subjects for HI Antibodies
Description: as for outcome 21
Time Frame: At Day 0 (PRE) and at Day 182
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity at Day 182, which included all evaluable subjects who met all eligibility criteria, who complied with the protocol requirements and for whom immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 54 | 84 | 47 | 52
Participants
  Flu A/CAL/7/09, PRE: number analyzed (Participants) | 54 | 82 | 47 | 52
  Flu A/CAL/7/09, PRE | 13 | 18 | 13 | 12
  Flu A/CAL/7/09, D182 | 54 | 84 | 45 | 50

27. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the Flu A/CAL/7/09 Influenza Strain - Preliminary Analysis
Description: Titers are presented as geometric mean titers (GMTs) and measured in titers.
Time Frame: At Day 0 (PRE) and at Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 66 | 59 | 61 | 62
Titers
  Flu A/CAL/7/09, PRE | 10.3 [7.4 to 14.5] | 6.2 [4.9 to 7.7] | 9.8 [6.9 to 13.9] | 10.9 [7.6 to 15.7]
  Flu A/CAL/7/09, D21: number analyzed (Participants) | 63 | 56 | 59 | 60
  Flu A/CAL/7/09, D21 | 387.9 [286.7 to 524.8] | 253.0 [185.8 to 344.4] | 141.4 [90.8 to 220.1] | 82.7 [52.9 to 129.5]

28. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the Flu A/CAL/7/09 Influenza Strain - First Analysis
Description: Titers are presented as geometric mean titers (GMTs) and measured in titers.
Time Frame: At Day 0 (PRE) and at Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 57 | 49 | 55 | 58
Titers
  Flu A/CAL/7/09, PRE | 10.8 [7.4 to 15.6] | 6.1 [4.7 to 7.8] | 10.5 [7.2 to 15.5] | 10.9 [7.5 to 15.8]
  Flu A/CAL/7/09, D21: number analyzed (Participants) | 57 | 49 | 55 | 57
  Flu A/CAL/7/09, D21 | 386.4 [280.3 to 532.6] | 270.1 [194.2 to 375.5] | 138.4 [86.3 to 222.0] | 83.4 [52.9 to 131.4]

29. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the Flu A/CAL/7/09 Influenza Strain - Second Analysis
Description: Titers are presented as geometric mean titers (GMTs) and measured in titers.
Time Frame: At Day 0 (PRE) and at Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 59 | 103 | 54 | 58
Titers
  Flu A/CAL/7/09, PRE: number analyzed (Participants) | 59 | 102 | 54 | 58
  Flu A/CAL/7/09, PRE | 10.5 [7.3 to 15.1] | 10.8 [8.2 to 14.3] | 10.7 [7.2 to 15.8] | 10.9 [7.5 to 15.8]
  Flu A/CAL/7/09, D21: number analyzed (Participants) | 59 | 103 | 54 | 57
  Flu A/CAL/7/09, D21 | 379.4 [277.9 to 518.0] | 377.3 [299.6 to 475.3] | 147.2 [92.4 to 234.3] | 83.4 [52.9 to 131.4]

30. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the Flu A/CAL/7/09 Influenza Strain - First Analysis
Description: Titers are presented as geometric mean titers (GMTs) and measured in titers.
Time Frame: At Day 0 (PRE) and at Day 42
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 43 | 42 | 46 | 44
Titers
  Flu A/CAL/7/09, PRE: number analyzed (Participants) | 43 | 40 | 46 | 44
  Flu A/CAL/7/09, PRE | 9.3 [6.4 to 13.5] | 5.7 [4.6 to 7.1] | 9.3 [6.4 to 13.6] | 9.5 [6.4 to 14.0]
  Flu A/CAL/7/09, D42 | 1444.4 [1146.0 to 1820.6] | 1238.5 [1050.2 to 1460.5] | 413.5 [296.6 to 576.4] | 228.0 [156.9 to 331.3]

31. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the Flu A/CAL/7/09 Influenza Strain - Second Analysis
Description: Titers are presented as geometric mean titers (GMTs) and measured in titers.
Time Frame: At Day 0 (PRE) and at Day 42
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 44 | 87 | 46 | 44
Titers
  Flu A/CAL/7/09, PRE: number analyzed (Participants) | 44 | 84 | 46 | 44
  Flu A/CAL/7/09, PRE | 9.2 [6.3 to 13.2] | 11.1 [8.2 to 15.1] | 9.3 [6.4 to 13.6] | 9.5 [6.4 to 14.0]
  Flu A/CAL/7/09, D42 | 1440.5 [1149.0 to 1805.8] | 1671.6 [1471.8 to 1898.4] | 413.5 [296.6 to 576.4] | 228.0 [156.9 to 331.3]

32. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the Flu A/CAL/7/09 Influenza Strain
Description: Titers are presented as geometric mean titers (GMTs) and measured in titers.
Time Frame: At Day 0 (PRE) and at Day 182
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 54 | 84 | 47 | 52
Titers
  Flu A/CAL/7/09, PRE: number analyzed (Participants) | 54 | 82 | 47 | 52
  Flu A/CAL/7/09, PRE | 9.6 [6.8 to 13.5] | 10.0 [7.3 to 13.6] | 11.9 [7.7 to 18.6] | 10.6 [7.2 to 15.7]
  Flu A/CAL/7/09, D182 | 296.2 [230.5 to 380.8] | 267.9 [219.5 to 327.0] | 122.7 [86.4 to 174.3] | 82.8 [59.5 to 115.2]

33. Secondary Outcome: Number of Seroconverted Subjects Against Flu A/CAL/7/09 Influenza Strain
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination reciprocal hemagglutination inhibition (HI) titer lower than (<) 10 and a post-vaccination reciprocal titer higher than or equal to (≥) 40, or a pre-vaccination reciprocal hemagglutination inhibition (HI) titer ≥ 10 and at least a 4-fold increase in post vaccination reciprocal titer against the vaccine virus.
Time Frame: At Day 182
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 54 | 82 | 47 | 52
Participants | 50 | 78 | 35 | 34

34. Secondary Outcome: Number of Seroprotected Subjects Against Flu A/CAL/7/09 Influenza Strain
Description: as for outcome 6
Time Frame: At Day 0 (PRE) and at Day 182
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 54 | 84 | 47 | 52
Participants
  Flu A/CAL/7/09, PRE: number analyzed (Participants) | 54 | 82 | 47 | 52
  Flu A/CAL/7/09, PRE | 10 | 16 | 12 | 12
  Flu A/CAL/7/09, D182 | 53 | 84 | 43 | 43

35. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against Flu A/CAL/7/09 Influenza Strain
Description: as for outcome 16
Time Frame: At Day 182
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 54 | 82 | 47 | 52
Fold change | 31.0 [22.7 to 42.4] | 26.6 [20.6 to 34.3] | 10.3 [7.1 to 14.8] | 7.8 [5.5 to 10.9]

36. Secondary Outcome: Number of Seropositive Subjects for Neutralizing Antibodies Against Flu A/Neth/602/09 Influenza Strain
Description: A seropositive subject was defined as a subject with antibody titers greater than or equal to (≥) 1:8. The vaccine strain assessed was Flu A/Neth/602/09 H1N1.
Time Frame: At Day 0 (PRE) and at Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 52 | 84 | 44 | 55
Participants
  Flu A/Neth/602/09, PRE: number analyzed (Participants) | 52 | 84 | 42 | 55
  Flu A/Neth/602/09, PRE | 25 | 30 | 17 | 20
  Flu A/Neth/602/09, D21: number analyzed (Participants) | 51 | 82 | 44 | 43
  Flu A/Neth/602/09, D21 | 51 | 82 | 39 | 35

37. Secondary Outcome: Titers for Neutralizing Antibodies Against the Flu A/Neth/602/09 Influenza Strain
Description: Titers are presented as geometric mean titers (GMTs) and measured in titers.
Time Frame: At Day 0 (PRE) and at Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 52 | 84 | 44 | 55
Titers
  Flu A/Neth/602/09, PRE: number analyzed (Participants) | 52 | 84 | 42 | 55
  Flu A/Neth/602/09, PRE | 19.3 [11.1 to 33.5] | 13.8 [9.0 to 20.9] | 15.0 [8.2 to 27.2] | 15.3 [8.8 to 26.6]
  Flu A/Neth/602/09, D21: number analyzed (Participants) | 51 | 82 | 44 | 43
  Flu A/Neth/602/09, D21 | 427.6 [244.5 to 748.0] | 296.1 [181.7 to 482.7] | 231.1 [111.9 to 477.3] | 138.3 [63.2 to 302.7]

38. Secondary Outcome: Number of Seropositive Subjects for Neutralizing Antibodies Against Flu A/Neth/602/09 Influenza Strain
Description: as for outcome 36
Time Frame: At Day 0 (PRE) and at Day 42
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 40 | 68 | 36 | 42
Participants
  Flu A/Neth/602/09, PRE: number analyzed (Participants) | 40 | 68 | 34 | 42
  Flu A/Neth/602/09, PRE | 18 | 26 | 13 | 13
  Flu A/Neth/602/09, D42: number analyzed (Participants) | 34 | 63 | 36 | 36
  Flu A/Neth/602/09, D42 | 34 | 63 | 35 | 33

39. Secondary Outcome: Titers for Neutralizing Antibodies Against the Flu A/Neth/602/09 Influenza Strain
Description: Titers are presented as geometric mean titers (GMTs) and measured in titers.
Time Frame: At Day 0 (PRE) and at Day 42
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 40 | 68 | 36 | 42
Titers
  Flu A/Neth/602/09, PRE: number analyzed (Participants) | 40 | 68 | 34 | 42
  Flu A/Neth/602/09, PRE | 16.7 [9.1 to 30.8] | 15.0 [9.3 to 24.1] | 12.0 [6.7 to 21.4] | 13.6 [7.3 to 25.5]
  Flu A/Neth/602/09, D42: number analyzed (Participants) | 34 | 63 | 36 | 36
  Flu A/Neth/602/09, D42 | 1389.3 [835.5 to 2310.4] | 1786.9 [1258.6 to 2537.0] | 428.4 [208.7 to 879.6] | 146.1 [74.3 to 287.5]

40. Secondary Outcome: Number of Subjects With Vaccine Responses for Neutralizing Antibody Concentrations
Description: Vaccine responses are defined as the incidence rate of vaccinated subjects with at least a 4-fold increase in post vaccination reciprocal titer relative to that prior to first vaccination. The vaccine strain assessed was Flu A/Neth/602/09 H1N1.
Time Frame: At Day 0 (PRE) and at Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 45 | 70 | 37 | 43
Participants | 41 | 57 | 27 | 24

41. Secondary Outcome: Number of Subjects With Vaccine Responses for Neutralizing Antibody Concentrations
Description: Vaccine response was defined as at least a 4-fold increase in post vaccination reciprocal titer relative to that prior to first vaccination. The vaccine strain assessed was Flu A/Neth/602/09.
Time Frame: At Day 0 (PRE) and at Day 42
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 32 | 54 | 30 | 34
Participants | 31 | 54 | 26 | 23

42. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms - Preliminary Analysis
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Arepanrix/F1 6M-5Y Group: Subjects, aged 6 months (M) - 5 years (Y), male or female, received 2 doses of Arepanrix™-formulation 1 (F1) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- Arepanrix/F1 6Y-9Y Group: Subjects, aged 6 years (Y) - 9 years, male or female, received 2 doses of Arepanrix™-formulation 1 (F1) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- Arepanrix/F2 6M-5Y Group: Subjects, aged 6 months (M) - 5 years (Y), male or female, received 2 doses of Arepanrix™-formulation 2 (F2) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- Arepanrix/F2 6Y-9Y Group: Subjects, aged 6 years (Y) - 9 years, male or female, received 2 doses of Arepanrix™-formulation 2 (F2) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- GSK2340273A/F1 6M-5Y Group: Subjects, aged 6 months (M) - 5 years (Y), male or female, received 2 doses of GSK2340273A-formulation 1 (F1) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- GSK2340273A/F1 6Y-9Y Group: Subjects, aged 6 years (Y) - 9 years, male or female, received 2 doses of GSK2340273A-formulation 1 (F1) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- GSK2340273A/F2 6M-5Y Group: Subjects, aged 6 months (M) - 5 years (Y), male or female, received 2 doses of GSK2340273A-formulation 2 (F2) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- GSK2340273A/F2 6Y-9Y Group: Subjects, aged 6 years (Y) - 9 years, male or female, received 2 doses of GSK2340273A-formulation 2 (F2) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
Arm/Group | Arepanrix/F1 6M-5Y Group | Arepanrix/F1 6Y-9Y Group | Arepanrix/F2 6M-5Y Group | Arepanrix/F2 6Y-9Y Group | GSK2340273A/F1 6M-5Y Group | GSK2340273A/F1 6Y-9Y Group | GSK2340273A/F2 6M-5Y Group | GSK2340273A/F2 6Y-9Y Group
Number analyzed (Participants) | 47 | 18 | 48 | 12 | 45 | 17 | 44 | 18
Participants
  Any Pain | 27 | 14 | 26 | 9 | 18 | 12 | 15 | 10
  Grade 3 Pain | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Any Redness | 5 | 4 | 4 | 2 | 1 | 0 | 1 | 1
  Grade 3 Redness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 0
  Grade 3 Swelling | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

43. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms - First Analysis
Description: as for outcome 42
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Arepanrix/F1 Out Group: Subjects, out of age interval, male or female, received 2 doses of Arepanrix™-formulation 1 (F1) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
Arm/Group | Arepanrix/F1 6M-5Y Group | Arepanrix/F1 6Y-9Y Group | Arepanrix/F1 Out Group | Arepanrix/F2 6M-5Y Group | Arepanrix/F2 6Y-9Y Group | GSK2340273A/F1 6M-5Y Group | GSK2340273A/F1 6Y-9Y Group | GSK2340273A/F2 6M-5Y Group | GSK2340273A/F2 6Y-9Y Group
Number analyzed (Participants) | 47 | 18 | 1 | 49 | 12 | 46 | 17 | 44 | 18
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 47 | 18 | 1 | 48 | 12 | 46 | 17 | 44 | 18
  Any Pain, Dose 1 | 27 | 14 | 1 | 26 | 9 | 19 | 12 | 15 | 10
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 47 | 18 | 1 | 48 | 12 | 46 | 17 | 44 | 18
  Grade 3 Pain, Dose 1 | 4 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Any Redness, Dose 1: number analyzed (Participants) | 47 | 18 | 1 | 48 | 12 | 46 | 17 | 44 | 18
  Any Redness, Dose 1 | 5 | 4 | 0 | 4 | 2 | 1 | 0 | 1 | 1
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 47 | 18 | 1 | 48 | 12 | 46 | 17 | 44 | 18
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 47 | 18 | 1 | 48 | 12 | 46 | 17 | 44 | 18
  Any Swelling, Dose 1 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 0
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 47 | 18 | 1 | 48 | 12 | 46 | 17 | 44 | 18
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 41 | 17 | 0 | 44 | 11 | 41 | 17 | 41 | 16
  Any Pain, Dose 2 | 22 | 13 | 0 | 25 | 7 | 11 | 8 | 9 | 7
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 41 | 17 | 0 | 44 | 11 | 41 | 17 | 41 | 16
  Grade 3 Pain, Dose 2 | 4 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 41 | 17 | 0 | 44 | 11 | 41 | 17 | 41 | 16
  Any Redness, Dose 2 | 5 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 41 | 17 | 0 | 44 | 11 | 41 | 17 | 41 | 16
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 41 | 17 | 0 | 44 | 11 | 41 | 17 | 41 | 16
  Any Swelling, Dose 2 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 41 | 17 | 0 | 44 | 11 | 41 | 17 | 41 | 16
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Across doses | 35 | 15 | 1 | 33 | 9 | 22 | 12 | 18 | 12
  Grade 3 Pain, Across doses | 7 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 1
  Any Redness, Across doses | 7 | 4 | 0 | 6 | 2 | 1 | 0 | 1 | 1
  Grade 3 Redness, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Across doses | 2 | 2 | 0 | 3 | 1 | 1 | 0 | 1 | 0
  Grade 3 Swelling, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

44. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms - Second Analysis
Description: as for outcome 42
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Arepanrix/F1 6M-35M Group: Subjects, aged 6 months (M) - 35 months, male or female, received 2 doses of Arepanrix™-formulation 1 (F1) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- Arepanrix/F1 3Y-5Y Group: Subjects, aged 3 years (Y) - 5 years, male or female, received 2 doses of Arepanrix™-formulation 1 (F1) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- Arepanrix/F2 6M-35M Group: Subjects, aged 6 months (M) - 35 months, male or female, received 2 doses of Arepanrix™-formulation 2 (F2) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- Arepanrix/F2 3Y-5Y Group: Subjects, aged 3 years (Y) - 5 years, male or female, received 2 doses of Arepanrix™-formulation 2 (F2) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- GSK2340273A/F1 6M-35M Group: Subjects, aged 6 months (M) - 35 months, male or female, received 2 doses of GSK2340273A-formulation 1 (F1) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- GSK2340273A/F1 3Y-5Y Group: Subjects, aged 3 years (Y) - 5 years, male or female, received 2 doses of GSK2340273A-formulation 1 (F1) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- GSK2340273A/F2 6M-35M Group: Subjects, aged 6 months (M) - 35 months, male or female, received 2 doses of GSK2340273A-formulation 2 (F2) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
- GSK2340273A/F2 3Y-6Y Group: Subjects, aged 3 years (Y) - 6 years, male or female, received 2 doses of GSK2340273A-formulation 2 (F2) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
Arm/Group | Arepanrix/F1 6M-35M Group | Arepanrix/F1 3Y-5Y Group | Arepanrix/F1 6Y-9Y Group | Arepanrix/F1 Out Group | Arepanrix/F2 6M-35M Group | Arepanrix/F2 3Y-5Y Group | Arepanrix/F2 6Y-9Y Group | GSK2340273A/F1 6M-35M Group | GSK2340273A/F1 3Y-5Y Group | GSK2340273A/F1 6Y-9Y Group | GSK2340273A/F2 6M-35M Group | GSK2340273A/F2 3Y-6Y Group | GSK2340273A/F2 6Y-9Y Group
Number analyzed (Participants) | 22 | 25 | 18 | 1 | 46 | 53 | 26 | 24 | 22 | 17 | 23 | 21 | 18
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 22 | 25 | 18 | 1 | 46 | 52 | 26 | 24 | 22 | 17 | 23 | 21 | 18
  Any Pain, Dose 1 | 12 | 15 | 14 | 1 | 20 | 34 | 22 | 10 | 9 | 12 | 8 | 7 | 10
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 22 | 25 | 18 | 1 | 46 | 52 | 26 | 24 | 22 | 17 | 23 | 21 | 18
  Grade 3 Pain, Dose 1 | 2 | 2 | 1 | 0 | 1 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 0
  Any Redness, Dose 1: number analyzed (Participants) | 22 | 25 | 18 | 1 | 46 | 52 | 26 | 24 | 22 | 17 | 23 | 21 | 18
  Any Redness, Dose 1 | 2 | 3 | 4 | 0 | 4 | 4 | 2 | 1 | 0 | 0 | 0 | 1 | 1
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 22 | 25 | 18 | 1 | 46 | 52 | 26 | 24 | 22 | 17 | 23 | 21 | 18
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 22 | 25 | 18 | 1 | 46 | 52 | 26 | 24 | 22 | 17 | 23 | 21 | 18
  Any Swelling, Dose 1 | 0 | 1 | 2 | 0 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 22 | 25 | 18 | 1 | 46 | 52 | 26 | 24 | 22 | 17 | 23 | 21 | 18
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 21 | 20 | 17 | 0 | 41 | 49 | 24 | 21 | 20 | 17 | 20 | 21 | 16
  Any Pain, Dose 2 | 12 | 10 | 13 | 0 | 18 | 35 | 19 | 5 | 6 | 8 | 4 | 5 | 7
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 21 | 20 | 17 | 0 | 41 | 49 | 24 | 21 | 20 | 17 | 20 | 21 | 16
  Grade 3 Pain, Dose 2 | 3 | 1 | 0 | 0 | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 21 | 20 | 17 | 0 | 41 | 49 | 24 | 21 | 20 | 17 | 20 | 21 | 16
  Any Redness, Dose 2 | 2 | 3 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 21 | 20 | 17 | 0 | 41 | 49 | 24 | 21 | 20 | 17 | 20 | 21 | 16
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 21 | 20 | 17 | 0 | 41 | 49 | 24 | 21 | 20 | 17 | 20 | 21 | 16
  Any Swelling, Dose 2 | 0 | 1 | 1 | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 21 | 20 | 17 | 0 | 41 | 49 | 24 | 21 | 20 | 17 | 20 | 21 | 16
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Across Doses | 16 | 19 | 15 | 1 | 25 | 44 | 22 | 11 | 11 | 12 | 9 | 9 | 12
  Grade 3 Pain, Across Doses | 4 | 3 | 1 | 0 | 3 | 5 | 5 | 1 | 0 | 1 | 0 | 0 | 1
  Any Redness, Across Doses | 3 | 4 | 4 | 0 | 5 | 5 | 2 | 1 | 0 | 0 | 0 | 1 | 1
  Grade 3 Redness, Across Doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Across Doses | 0 | 2 | 2 | 0 | 4 | 4 | 3 | 1 | 0 | 0 | 0 | 1 | 0
  Grade 3 Swelling, Across Doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

45. Secondary Outcome: Number of Subjects Less Than 6 Years Old With Any, Grade 3 and Related Solicited General Symptoms - Preliminary Analysis
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and temperature [defined as axillary temperature equal to or above (≥) 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 loss of appetite= not eating at all. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 6M-5Y Group | Arepanrix/F2 6M-5Y Group | GSK2340273A/F1 6M-5Y Group | GSK2340273A/F2 6M-5Y Group
Number analyzed (Participants) | 47 | 48 | 45 | 44
Participants
  Any Drowsiness | 11 | 11 | 8 | 9
  Grade 3 Drowsiness | 2 | 1 | 0 | 0
  Related Drowsiness | 5 | 8 | 5 | 7
  Any Irritability | 22 | 18 | 14 | 8
  Grade 3 Irritability | 3 | 3 | 0 | 0
  Related Irritability | 19 | 15 | 12 | 8
  Any Loss of appetite | 16 | 17 | 6 | 9
  Grade 3 Loss of appetite | 1 | 1 | 0 | 1
  Related Loss of appetite | 9 | 12 | 3 | 8
  Any Temperature (Axillary) | 8 | 6 | 2 | 1
  Grade 3 Temperature (Axillary) | 1 | 0 | 0 | 0
  Related Temperature (Axillary) | 6 | 3 | 1 | 1

46. Secondary Outcome: Number of Subjects Aged Between 6 to Less Than 9 Years With Any, Grade 3 and Related Solicited General Symptoms - Preliminary Analysis
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache, joint pain at other location, muscle aches, shivering, sweating, temperature [defined as axillary temperature equal to or above (≥) 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 6Y-9Y Group | Arepanrix/F2 6Y-9Y Group | GSK2340273A/F1 6Y-9Y Group | GSK2340273A/F2 6Y-9Y Group
Number analyzed (Participants) | 18 | 12 | 17 | 18
Participants
  Any Fatigue | 3 | 4 | 4 | 4
  Grade 3 Fatigue | 0 | 0 | 1 | 0
  Related Fatigue | 2 | 3 | 4 | 3
  Any Gastro-intestinal symptoms | 1 | 2 | 3 | 2
  Grade 3 Gastro-intestinal symptoms | 0 | 0 | 0 | 0
  Related Gastro-intestinal symptoms | 0 | 1 | 3 | 0
  Any Headache | 4 | 4 | 2 | 2
  Grade 3 Headache | 0 | 0 | 0 | 0
  Related Headache | 3 | 2 | 1 | 2
  Any Joint pain at other location | 0 | 0 | 2 | 1
  Grade 3 Joint pain at other location | 0 | 0 | 0 | 0
  Related Joint pain at other location | 0 | 0 | 2 | 0
  Any Muscle aches | 4 | 2 | 3 | 1
  Grade 3 Muscle aches | 0 | 0 | 0 | 0
  Related Muscle aches | 4 | 2 | 3 | 1
  Any Shivering | 0 | 0 | 1 | 0
  Grade 3 Shivering | 0 | 0 | 0 | 0
  Related Shivering | 0 | 0 | 1 | 0
  Any Sweating | 1 | 1 | 2 | 1
  Grade 3 Sweating | 0 | 0 | 0 | 0
  Related Sweating | 1 | 0 | 2 | 0
  Any Temperature (Axillary) | 4 | 2 | 1 | 0
  Grade 3 Temperature (Axillary) | 0 | 0 | 0 | 0
  Related Temperature (Axillary) | 3 | 2 | 1 | 0

47. Secondary Outcome: Number of Subjects Less Than 6 Years Old With Any, Grade 3 and Related Solicited General Symptoms - First Analysis
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and temperature [defined as axillary temperature equal to or above (≥) 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 6M-5Y Group | Arepanrix/F2 6M-5Y Group | GSK2340273A/F1 6M-5Y Group | GSK2340273A/F2 6M-5Y Group
Number analyzed (Participants) | 47 | 49 | 46 | 44
Participants
  Any Drowsiness, Dose 1: number analyzed (Participants) | 47 | 48 | 46 | 44
  Any Drowsiness, Dose 1 | 11 | 11 | 8 | 9
  Grade 3 Drowsiness, Dose 1: number analyzed (Participants) | 47 | 48 | 46 | 44
  Grade 3 Drowsiness, Dose 1 | 2 | 1 | 0 | 0
  Related Drowsiness, Dose 1: number analyzed (Participants) | 47 | 48 | 46 | 44
  Related Drowsiness, Dose 1 | 5 | 8 | 5 | 7
  Any Irritability, Dose 1: number analyzed (Participants) | 47 | 48 | 46 | 44
  Any Irritability, Dose 1 | 22 | 18 | 15 | 8
  Grade 3 Irritability, Dose 1: number analyzed (Participants) | 47 | 48 | 46 | 44
  Grade 3 Irritability, Dose 1 | 3 | 3 | 1 | 0
  Related Irritability, Dose 1: number analyzed (Participants) | 47 | 48 | 46 | 44
  Related Irritability, Dose 1 | 19 | 15 | 12 | 8
  Any Loss of appetite, Dose 1: number analyzed (Participants) | 47 | 48 | 46 | 44
  Any Loss of appetite, Dose 1 | 16 | 17 | 6 | 9
  Grade 3 Loss of appetite, Dose 1: number analyzed (Participants) | 47 | 48 | 46 | 44
  Grade 3 Loss of appetite, Dose 1 | 1 | 1 | 0 | 1
  Related Loss of appetite, Dose 1: number analyzed (Participants) | 47 | 48 | 46 | 44
  Related Loss of appetite, Dose 1 | 9 | 12 | 3 | 8
  Any Temperature (Axillary), Dose 1: number analyzed (Participants) | 47 | 48 | 46 | 44
  Any Temperature (Axillary), Dose 1 | 9 | 6 | 2 | 1
  Grade 3 Temperature (Axillary), Dose 1: number analyzed (Participants) | 47 | 48 | 46 | 44
  Grade 3 Temperature (Axillary), Dose 1 | 1 | 0 | 0 | 0
  Related Temperature (Axillary), Dose 1: number analyzed (Participants) | 47 | 48 | 46 | 44
  Related Temperature (Axillary), Dose 1 | 8 | 3 | 1 | 1
  Any Drowsiness, Dose 2: number analyzed (Participants) | 41 | 44 | 41 | 41
  Any Drowsiness, Dose 2 | 13 | 6 | 7 | 7
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 41 | 44 | 41 | 41
  Grade 3 Drowsiness, Dose 2 | 5 | 0 | 0 | 0
  Related Drowsiness, Dose 2: number analyzed (Participants) | 41 | 44 | 41 | 41
  Related Drowsiness, Dose 2 | 9 | 2 | 5 | 7
  Any Irritability, Dose 2: number analyzed (Participants) | 41 | 44 | 41 | 41
  Any Irritability, Dose 2 | 19 | 12 | 13 | 11
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 41 | 44 | 41 | 41
  Grade 3 Irritability, Dose 2 | 3 | 1 | 2 | 2
  Related Irritability, Dose 2: number analyzed (Participants) | 41 | 44 | 41 | 41
  Related Irritability, Dose 2 | 18 | 11 | 12 | 11
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 41 | 44 | 41 | 41
  Any Loss of appetite, Dose 2 | 18 | 10 | 7 | 5
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 41 | 44 | 41 | 41
  Grade 3 Loss of appetite, Dose 2 | 1 | 2 | 0 | 0
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 41 | 44 | 41 | 41
  Related Loss of appetite, Dose 2 | 15 | 8 | 5 | 5
  Any Temperature (Axillary), Dose 2: number analyzed (Participants) | 41 | 44 | 41 | 41
  Any Temperature (Axillary), Dose 2 | 13 | 7 | 3 | 3
  Grade 3 Temperature (Axillary), Dose 2: number analyzed (Participants) | 41 | 44 | 41 | 41
  Grade 3 Temperature (Axillary), Dose 2 | 5 | 0 | 0 | 0
  Related Temperature (Axillary), Dose 2: number analyzed (Participants) | 41 | 44 | 41 | 41
  Related Temperature (Axillary), Dose 2 | 11 | 6 | 2 | 0
  Any Drowsiness, Across doses | 17 | 15 | 13 | 14
  Grade 3 Drowsiness, Across doses | 6 | 1 | 0 | 0
  Related Drowsiness, Across doses | 10 | 9 | 9 | 12
  Any Irritability, Across doses | 28 | 22 | 21 | 17
  Grade 3 Irritability, Across doses | 6 | 4 | 3 | 2
  Related Irritability, Across doses | 25 | 20 | 17 | 17
  Any Loss of appetite, Across doses | 25 | 23 | 11 | 11
  Grade 3 Loss of appetite, Across doses | 2 | 3 | 0 | 1
  Related Loss of appetite, Across doses | 17 | 17 | 7 | 10
  Any Temperature (Axillary), Across doses | 19 | 11 | 4 | 4
  Grade 3 Temperature (Axillary), Across doses | 6 | 0 | 0 | 0
  Related Temperature (Axillary), Across doses | 16 | 8 | 2 | 1

48. Secondary Outcome: Number of Subjects Aged Between 6 to Less Than 9 Years With Any, Grade 3 and Related Solicited General Symptoms - First Analysis
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache, joint pain at other location, muscle aches, and shivering, sweating, temperature [defined as axillary temperature equal to or above (≥) 38 degrees Celsius (° C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 6Y-9Y Group | Arepanrix/F2 6Y-9Y Group | GSK2340273A/F1 6Y-9Y Group | GSK2340273A/F2 6Y-9Y Group
Number analyzed (Participants) | 18 | 12 | 17 | 18
Participants
  Any Fatigue, Dose 1 | 3 | 4 | 4 | 4
  Grade 3 Fatigue, Dose 1 | 0 | 0 | 1 | 0
  Related Fatigue, Dose 1 | 2 | 3 | 4 | 3
  Any Gastrointestinal symptoms, Dose 1 | 1 | 2 | 3 | 2
  Grade 3 Gastrointestinal symptoms, Dose 1 | 0 | 0 | 1 | 0
  Related Gastrointestinal symptoms, Dose 1 | 0 | 1 | 3 | 0
  Any Headache, Dose 1 | 4 | 4 | 2 | 2
  Grade 3 Headache, Dose 1 | 0 | 0 | 0 | 0
  Related Headache, Dose 1 | 3 | 2 | 1 | 2
  Any Joint pain at other location, Dose 1 | 0 | 0 | 2 | 1
  Grade 3 Joint pain at other location, Dose 1 | 0 | 0 | 0 | 0
  Related Joint pain at other location, Dose 1 | 0 | 0 | 2 | 0
  Any Muscle aches, Dose 1 | 4 | 2 | 3 | 1
  Grade 3 Muscle aches, Dose 1 | 0 | 0 | 0 | 0
  Related Muscle aches, Dose 1 | 4 | 2 | 3 | 1
  Any Shivering, Dose 1 | 0 | 0 | 1 | 0
  Grade 3 Shivering, Dose 1 | 0 | 0 | 0 | 0
  Related Shivering, Dose 1 | 0 | 0 | 1 | 0
  Any Sweating, Dose 1 | 1 | 1 | 2 | 1
  Grade 3 Sweating, Dose 1 | 0 | 0 | 0 | 0
  Related Sweating, Dose 1 | 1 | 0 | 2 | 0
  Any Temperature (Axillary), Dose 1 | 5 | 2 | 1 | 0
  Grade 3 Temperature (Axillary), Dose 1 | 0 | 0 | 0 | 0
  Related Temperature (Axillary), Dose 1 | 3 | 2 | 1 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Any Fatigue, Dose 2 | 3 | 3 | 3 | 4
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Grade 3 Fatigue, Dose 2 | 0 | 1 | 0 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Related Fatigue, Dose 2 | 3 | 2 | 3 | 3
  Any Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Any Gastrointestinal symptoms, Dose 2 | 0 | 2 | 1 | 5
  Grade 3 Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Grade 3 Gastrointestinal symptoms, Dose 2 | 0 | 0 | 0 | 1
  Related Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Related Gastrointestinal symptoms, Dose 2 | 0 | 2 | 1 | 4
  Any Headache, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Any Headache, Dose 2 | 8 | 3 | 2 | 4
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Grade 3 Headache, Dose 2 | 0 | 0 | 0 | 1
  Related Headache, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Related Headache, Dose 2 | 8 | 3 | 2 | 3
  Any Joint pain at other location, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Any Joint pain at other location, Dose 2 | 2 | 4 | 0 | 1
  Grade 3 Joint pain at other location, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Grade 3 Joint pain at other location, Dose 2 | 0 | 1 | 0 | 0
  Related Joint pain at other location, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Related Joint pain at other location, Dose 2 | 2 | 4 | 0 | 0
  Any Muscle aches, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Any Muscle aches, Dose 2 | 7 | 2 | 1 | 2
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Grade 3 Muscle aches, Dose 2 | 0 | 1 | 0 | 0
  Related Muscle aches, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Related Muscle aches, Dose 2 | 7 | 2 | 1 | 1
  Any Shivering, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Any Shivering, Dose 2 | 4 | 2 | 2 | 1
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Grade 3 Shivering, Dose 2 | 0 | 0 | 0 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Related Shivering, Dose 2 | 4 | 2 | 2 | 0
  Any Sweating, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Any Sweating, Dose 2 | 1 | 1 | 0 | 2
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Grade 3 Sweating, Dose 2 | 0 | 0 | 0 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Related Sweating, Dose 2 | 1 | 1 | 0 | 1
  Any Temperature (Axillary), Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Any Temperature (Axillary), Dose 2 | 5 | 2 | 0 | 2
  Grade 3 Temperature (Axillary), Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Grade 3 Temperature (Axillary), Dose 2 | 2 | 0 | 0 | 0
  Related Temperature (Axillary), Dose 2: number analyzed (Participants) | 17 | 11 | 17 | 16
  Related Temperature (Axillary), Dose 2 | 5 | 2 | 0 | 1
  Any Fatigue, Across doses | 6 | 5 | 4 | 8
  Grade 3 Fatigue, Across doses | 0 | 1 | 1 | 0
  Related Fatigue, Across doses | 5 | 4 | 4 | 6
  Any Gastrointestinal symptoms, Across doses | 1 | 3 | 3 | 7
  Grade 3 Gastrointestinal symptoms, Across doses | 0 | 0 | 1 | 1
  Related Gastrointestinal symptoms, Across doses | 0 | 3 | 3 | 4
  Any Headache, Across doses | 9 | 5 | 4 | 5
  Grade 3 Headache, Across doses | 0 | 0 | 0 | 1
  Related Headache, Across doses | 9 | 4 | 3 | 4
  Any Joint pain at other location, Across doses | 2 | 4 | 2 | 2
  Grade 3 Joint pain at other location, Across doses | 0 | 1 | 0 | 0
  Related Joint pain at other location, Across doses | 2 | 4 | 2 | 0
  Any Muscle aches, Across doses | 8 | 3 | 3 | 3
  Grade 3 Muscle aches, Across doses | 0 | 1 | 0 | 0
  Related Muscle aches, Across doses | 8 | 3 | 3 | 2
  Any Shivering, Across doses | 4 | 2 | 2 | 1
  Grade 3 Shivering, Across doses | 0 | 0 | 0 | 0
  Related Shivering, Across doses | 4 | 2 | 2 | 0
  Any Sweating, Across doses | 2 | 1 | 2 | 3
  Grade 3 Sweating, Across doses | 0 | 0 | 0 | 0
  Related Sweating, Across doses | 2 | 1 | 2 | 1
  Any Temperature (Axillary), Across doses | 9 | 4 | 1 | 2
  Grade 3 Temperature (Axillary), Across doses | 2 | 0 | 0 | 0
  Related Temperature (Axillary), Across doses | 7 | 4 | 1 | 1

49. Secondary Outcome: Number of Subjects Less Than 6 Years Old With Any, Grade 3 and Related Solicited General Symptoms - Second Analysis
Description: as for outcome 47
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340273A/F2 3Y-5Y Group: Subjects, aged 3 years (Y) - 5 years, male or female, received 2 doses of GSK2340273A-formulation 2 (F2) vaccine administered at a 21-day interval. The first dose was administered intramuscularly in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) or left anterolateral thigh (for children < 12 months of age). The second vaccine dose was administered in the deltoid region of the dominant arm (or right arm) or right anterolateral thigh (children < 12 months of age).
Arm/Group | Arepanrix/F1 6M-35M Group | Arepanrix/F1 3Y-5Y Group | Arepanrix/F2 6M-35M Group | Arepanrix/F2 3Y-5Y Group | GSK2340273A/F1 6M-35M Group | GSK2340273A/F1 3Y-5Y Group | GSK2340273A/F2 6M-35M Group | GSK2340273A/F2 3Y-5Y Group
Number analyzed (Participants) | 22 | 25 | 46 | 53 | 24 | 22 | 23 | 21
Participants
  Any Drowsiness, Dose 1: number analyzed (Participants) | 22 | 25 | 46 | 52 | 24 | 22 | 23 | 21
  Any Drowsiness, Dose 1 | 6 | 5 | 20 | 13 | 4 | 4 | 6 | 3
  Grade 3 Drowsiness, Dose 1: number analyzed (Participants) | 22 | 25 | 46 | 52 | 24 | 22 | 23 | 21
  Grade 3 Drowsiness, Dose 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
  Related Drowsiness, Dose 1: number analyzed (Participants) | 22 | 25 | 46 | 52 | 24 | 22 | 23 | 21
  Related Drowsiness, Dose 1 | 3 | 2 | 13 | 4 | 3 | 2 | 5 | 2
  Any Irritability, Dose 1: number analyzed (Participants) | 22 | 25 | 46 | 52 | 24 | 22 | 23 | 21
  Any Irritability, Dose 1 | 14 | 8 | 22 | 14 | 9 | 6 | 8 | 0
  Grade 3 Irritability, Dose 1: number analyzed (Participants) | 22 | 25 | 46 | 52 | 24 | 22 | 23 | 21
  Grade 3 Irritability, Dose 1 | 1 | 2 | 6 | 0 | 1 | 0 | 0 | 0
  Related Irritability, Dose 1: number analyzed (Participants) | 22 | 25 | 46 | 52 | 24 | 22 | 23 | 21
  Related Irritability, Dose 1 | 13 | 6 | 15 | 8 | 8 | 4 | 8 | 0
  Any Loss of appetite, Dose 1: number analyzed (Participants) | 22 | 25 | 46 | 52 | 24 | 22 | 23 | 21
  Any Loss of appetite, Dose 1 | 9 | 7 | 19 | 12 | 2 | 4 | 8 | 1
  Grade 3 Loss of appetite, Dose 1: number analyzed (Participants) | 22 | 25 | 46 | 52 | 24 | 22 | 23 | 21
  Grade 3 Loss of appetite, Dose 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0
  Related Loss of appetite, Dose 1: number analyzed (Participants) | 22 | 25 | 46 | 52 | 24 | 22 | 23 | 21
  Related Loss of appetite, Dose 1 | 6 | 3 | 12 | 5 | 1 | 2 | 7 | 1
  Any Temperature (Axillary), Dose 1: number analyzed (Participants) | 22 | 25 | 46 | 52 | 24 | 22 | 23 | 21
  Any Temperature (Axillary), Dose 1 | 5 | 4 | 6 | 9 | 0 | 2 | 0 | 1
  Grade 3 Temperature (Axillary), Dose 1: number analyzed (Participants) | 22 | 25 | 46 | 52 | 24 | 22 | 23 | 21
  Grade 3 Temperature (Axillary), Dose 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Temperature (Axillary), Dose 1: number analyzed (Participants) | 22 | 25 | 46 | 52 | 24 | 22 | 23 | 21
  Related Temperature (Axillary), Dose 1 | 4 | 4 | 1 | 2 | 0 | 1 | 0 | 1
  Any Drowsiness, Dose 2: number analyzed (Participants) | 21 | 20 | 41 | 49 | 21 | 20 | 20 | 21
  Any Drowsiness, Dose 2 | 8 | 5 | 9 | 9 | 5 | 2 | 5 | 2
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 21 | 20 | 41 | 49 | 21 | 20 | 20 | 21
  Grade 3 Drowsiness, Dose 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Related Drowsiness, Dose 2: number analyzed (Participants) | 21 | 20 | 41 | 49 | 21 | 20 | 20 | 21
  Related Drowsiness, Dose 2 | 7 | 2 | 5 | 5 | 4 | 1 | 5 | 2
  Any Irritability, Dose 2: number analyzed (Participants) | 21 | 20 | 41 | 49 | 21 | 20 | 20 | 21
  Any Irritability, Dose 2 | 13 | 6 | 23 | 10 | 10 | 3 | 6 | 5
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 21 | 20 | 41 | 49 | 21 | 20 | 20 | 21
  Grade 3 Irritability, Dose 2 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 1
  Related Irritability, Dose 2: number analyzed (Participants) | 21 | 20 | 41 | 49 | 21 | 20 | 20 | 21
  Related Irritability, Dose 2 | 13 | 5 | 19 | 8 | 9 | 3 | 6 | 5
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 21 | 20 | 41 | 49 | 21 | 20 | 20 | 21
  Any Loss of appetite, Dose 2 | 11 | 7 | 13 | 10 | 7 | 0 | 4 | 1
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 21 | 20 | 41 | 49 | 21 | 20 | 20 | 21
  Grade 3 Loss of appetite, Dose 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 21 | 20 | 41 | 49 | 21 | 20 | 20 | 21
  Related Loss of appetite, Dose 2 | 11 | 4 | 10 | 7 | 5 | 0 | 4 | 1
  Any Temperature (Axillary), Dose 2: number analyzed (Participants) | 21 | 20 | 41 | 49 | 21 | 20 | 20 | 21
  Any Temperature (Axillary), Dose 2 | 10 | 3 | 6 | 8 | 2 | 1 | 1 | 2
  Grade 3 Temperature (Axillary), Dose 2: number analyzed (Participants) | 21 | 20 | 41 | 49 | 21 | 20 | 20 | 21
  Grade 3 Temperature (Axillary), Dose 2 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Related Temperature (Axillary), Dose 2: number analyzed (Participants) | 21 | 20 | 41 | 49 | 21 | 20 | 20 | 21
  Related Temperature (Axillary), Dose 2 | 9 | 2 | 5 | 5 | 1 | 1 | 0 | 0
  Any Drowsiness, Across doses | 10 | 7 | 23 | 19 | 7 | 6 | 9 | 5
  Grade 3 Drowsiness, Across doses | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 0
  Related Drowsiness, Across doses | 7 | 3 | 16 | 7 | 6 | 3 | 8 | 4
  Any Irritability, Across doses | 19 | 9 | 30 | 20 | 14 | 7 | 12 | 5
  Grade 3 Irritability, Across doses | 3 | 3 | 7 | 0 | 2 | 1 | 1 | 1
  Related Irritability, Across doses | 18 | 7 | 23 | 14 | 12 | 5 | 12 | 5
  Any Loss of appetite, Across doses | 15 | 10 | 26 | 19 | 7 | 4 | 9 | 2
  Grade 3 Loss of appetite, Across doses | 1 | 1 | 3 | 2 | 0 | 0 | 1 | 0
  Related Loss of appetite, Across doses | 12 | 5 | 19 | 10 | 5 | 2 | 8 | 2
  Any Temperature (Axillary), Across doses | 13 | 6 | 10 | 14 | 2 | 2 | 1 | 3
  Grade 3 Temperature (Axillary), Across doses | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Related Temperature (Axillary), Across doses | 11 | 5 | 6 | 6 | 1 | 1 | 0 | 1

50. Secondary Outcome: Number of Subjects Aged Between 6 and 9 Years With Any, Grade 3 and Related Solicited General Symptoms- Second Analysis
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache, joint pain at other location, muscle aches, shivering, sweating and temperature [defined as axillary temperature equal to or above (≥) 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 6Y-9Y Group | Arepanrix/F2 6Y-9Y Group | GSK2340273A/F1 6Y-9Y Group | GSK2340273A/F2 6Y-9Y Group
Number analyzed (Participants) | 18 | 26 | 17 | 18
Participants
  Any Fatigue, Dose 1 | 3 | 8 | 4 | 4
  Grade 3 Fatigue, Dose 1 | 0 | 1 | 1 | 0
  Related Fatigue, Dose 1 | 2 | 4 | 4 | 3
  Any Gastrointestinal symptoms, Dose 1 | 1 | 4 | 3 | 2
  Grade 3 Gastrointestinal symptoms, Dose 1 | 0 | 1 | 1 | 0
  Related Gastrointestinal symptoms, Dose 1 | 0 | 1 | 3 | 0
  Any Headache, Dose 1 | 4 | 9 | 2 | 2
  Grade 3 Headache, Dose 1 | 0 | 1 | 0 | 0
  Related Headache, Dose 1 | 3 | 3 | 1 | 2
  Any Joint pain at other location, Dose 1 | 0 | 5 | 2 | 1
  Grade 3 Joint pain at other location, Dose 1 | 0 | 1 | 0 | 0
  Related Joint pain at other location, Dose 1 | 0 | 1 | 2 | 0
  Any Muscle aches, Dose 1 | 4 | 7 | 3 | 1
  Grade 3 Muscle aches, Dose 1 | 0 | 1 | 0 | 0
  Related Muscle aches, Dose 1 | 4 | 5 | 3 | 1
  Any Shivering, Dose 1 | 0 | 2 | 1 | 0
  Grade 3 Shivering, Dose 1 | 0 | 0 | 0 | 0
  Related Shivering, Dose 1 | 0 | 0 | 1 | 0
  Any Sweating, Dose 1 | 1 | 2 | 2 | 1
  Grade 3 Sweating, Dose 1 | 0 | 0 | 0 | 0
  Related Sweating, Dose 1 | 1 | 0 | 2 | 0
  Any Temperature (Axillary), Dose 1 | 5 | 6 | 1 | 0
  Grade 3 Temperature (Axillary), Dose 1 | 0 | 0 | 0 | 0
  Related Temperature (Axillary), Dose 1 | 3 | 2 | 1 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Any Fatigue, Dose 2 | 3 | 7 | 3 | 4
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Grade 3 Fatigue, Dose 2 | 0 | 2 | 0 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Related Fatigue, Dose 2 | 3 | 3 | 3 | 3
  Any Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Any Gastrointestinal symptoms, Dose 2 | 0 | 6 | 1 | 5
  Grade 3 Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Grade 3 Gastrointestinal symptoms, Dose 2 | 0 | 1 | 0 | 1
  Related Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Related Gastrointestinal symptoms, Dose 2 | 0 | 2 | 1 | 4
  Any Headache, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Any Headache, Dose 2 | 8 | 7 | 2 | 4
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Grade 3 Headache, Dose 2 | 0 | 1 | 0 | 1
  Related Headache, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Related Headache, Dose 2 | 8 | 4 | 2 | 3
  Any Joint pain at other location, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Any Joint pain at other location, Dose 2 | 2 | 6 | 0 | 1
  Grade 3 Joint pain at other location, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Grade 3 Joint pain at other location, Dose 2 | 0 | 2 | 0 | 0
  Related Joint pain at other location, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Related Joint pain at other location, Dose 2 | 2 | 5 | 0 | 0
  Any Muscle aches, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Any Muscle aches, Dose 2 | 7 | 8 | 1 | 2
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Grade 3 Muscle aches, Dose 2 | 0 | 3 | 0 | 0
  Related Muscle aches, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Related Muscle aches, Dose 2 | 7 | 6 | 1 | 1
  Any Shivering, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Any Shivering, Dose 2 | 4 | 3 | 2 | 1
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Grade 3 Shivering, Dose 2 | 0 | 1 | 0 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Related Shivering, Dose 2 | 4 | 2 | 2 | 0
  Any Sweating, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Any Sweating, Dose 2 | 1 | 3 | 0 | 2
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Grade 3 Sweating, Dose 2 | 0 | 1 | 0 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Related Sweating, Dose 2 | 1 | 1 | 0 | 1
  Any Temperature (Axillary), Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Any Temperature (Axillary), Dose 2 | 5 | 6 | 0 | 2
  Grade 3 Temperature (Axillary), Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Grade 3 Temperature (Axillary), Dose 2 | 2 | 2 | 0 | 0
  Related Temperature (Axillary), Dose 2: number analyzed (Participants) | 17 | 24 | 17 | 16
  Related Temperature (Axillary), Dose 2 | 5 | 4 | 0 | 1
  Any Fatigue, Across doses | 6 | 11 | 4 | 8
  Grade 3 Fatigue, Across doses | 0 | 2 | 1 | 0
  Related Fatigue, Across doses | 5 | 6 | 4 | 6
  Any Gastrointestinal symptoms, Across doses | 1 | 8 | 3 | 7
  Grade 3 Gastrointestinal symptoms, Across doses | 0 | 1 | 1 | 1
  Related Gastrointestinal symptoms, Across doses | 0 | 3 | 3 | 4
  Any Headache, Across doses | 9 | 12 | 4 | 5
  Grade 3 Headache, Across doses | 0 | 1 | 0 | 1
  Related Headache, Across doses | 9 | 6 | 3 | 4
  Any Joint pain at other location, Across doses | 2 | 10 | 2 | 2
  Grade 3 Joint pain at other location, Across doses | 0 | 2 | 0 | 0
  Related Joint pain at other location, Across doses | 2 | 6 | 2 | 0
  Any Muscle aches, Across doses | 8 | 11 | 3 | 3
  Grade 3 Muscle aches, Across doses | 0 | 3 | 0 | 0
  Related Muscle aches, Across doses | 8 | 8 | 3 | 2
  Any Shivering, Across doses | 4 | 5 | 2 | 1
  Grade 3 Shivering, Across doses | 0 | 1 | 0 | 0
  Related Shivering, Across doses | 4 | 2 | 2 | 0
  Any Sweating, Across doses | 2 | 4 | 2 | 3
  Grade 3 Sweating, Across doses | 0 | 1 | 0 | 0
  Related Sweating, Across doses | 2 | 1 | 2 | 1
  Any Temperature (Axillary), Across doses | 9 | 9 | 1 | 2
  Grade 3 Temperature (Axillary), Across doses | 2 | 2 | 0 | 0
  Related Temperature (Axillary), Across doses | 7 | 6 | 1 | 1

51. Secondary Outcome: Number of Subjects With Haematological Laboratory Abnormalities - Preliminary Analysis
Description: Among haematological parameters assessed were basophils [BAS], eosinophils [EOS], hematocrit [HCT], hemoglobin level [HGB], lymphocytes [LYM], monocytes [MON], neutrophils [NEU], platelet count [PLC], red blood cells [RBC] and white blood cells [WBC]. Haematological laboratory values were unknown, below, within or above the laboratory reference range defined for the specified time point and laboratory parameter.
Time Frame: At Day 0 (PRE), at Day 7 and at Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 66 | 60 | 60 | 61
Participants
  BAS, PRE: number analyzed (Participants) | 37 | 37 | 28 | 28
  BAS, PRE: Unknown | 2 | 6 | 4 | 0
  BAS, PRE: Below | 0 | 0 | 0 | 0
  BAS, PRE: Within | 35 | 31 | 24 | 28
  BAS, PRE: Above | 0 | 0 | 0 | 0
  BAS, D7: Unknown | 5 | 4 | 4 | 3
  BAS, D7: Below | 0 | 0 | 0 | 0
  BAS, D7: Within | 61 | 56 | 56 | 58
  BAS, D7: Above | 0 | 0 | 0 | 0
  BAS, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  BAS, D21: Unknown | 1 | 3 | 6 | 0
  BAS, D21: Below | 0 | 0 | 0 | 0
  BAS, D21: Within | 64 | 54 | 52 | 61
  BAS, D21: Above | 0 | 0 | 0 | 0
  EOS, PRE: number analyzed (Participants) | 37 | 37 | 28 | 28
  EOS, PRE: Unknown | 2 | 6 | 4 | 0
  EOS, PRE: Below | 5 | 1 | 2 | 4
  EOS, PRE: Within | 28 | 28 | 20 | 20
  EOS, PRE: Above | 2 | 2 | 2 | 4
  EOS, D7: Unknown | 5 | 4 | 4 | 3
  EOS, D7: Below | 7 | 8 | 8 | 6
  EOS, D7: Within | 50 | 42 | 46 | 45
  EOS, D7: Above | 4 | 6 | 2 | 7
  EOS, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  EOS, D21: Unknown | 1 | 3 | 6 | 0
  EOS, D21: Below | 5 | 6 | 5 | 7
  EOS, D21: Within | 54 | 42 | 46 | 51
  EOS, D21: Above | 5 | 6 | 1 | 3
  HCT, PRE: number analyzed (Participants) | 37 | 37 | 28 | 28
  HCT, PRE: Unknown | 2 | 6 | 4 | 0
  HCT, PRE: Below | 2 | 3 | 0 | 3
  HCT, PRE: Within | 31 | 24 | 22 | 24
  HCT, PRE: Above | 2 | 4 | 2 | 1
  HCT, D7: Unknown | 5 | 4 | 4 | 3
  HCT, D7: Below | 6 | 7 | 4 | 6
  HCT, D7: Within | 52 | 47 | 48 | 49
  HCT, D7: Above | 3 | 2 | 4 | 3
  HCT, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  HCT, D21: Unknown | 1 | 3 | 6 | 0
  HCT, D21: Below | 7 | 10 | 7 | 7
  HCT, D21: Within | 54 | 41 | 42 | 53
  HCT, D21: Above | 3 | 3 | 3 | 1
  HGB, PRE: number analyzed (Participants) | 37 | 37 | 28 | 28
  HGB, PRE: Unknown | 2 | 6 | 4 | 0
  HGB, PRE: Below | 1 | 2 | 0 | 3
  HGB, PRE: Within | 31 | 25 | 22 | 23
  HGB, PRE: Above | 3 | 4 | 2 | 2
  HGB, D7: Unknown | 5 | 3 | 4 | 3
  HGB, D7: Below | 4 | 5 | 1 | 2
  HGB, D7: Within | 55 | 50 | 51 | 52
  HGB, D7: Above | 2 | 2 | 4 | 4
  HGB, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  HGB, D21: Unknown | 1 | 3 | 6 | 0
  HGB, D21: Below | 5 | 3 | 3 | 3
  HGB, D21: Within | 55 | 48 | 46 | 56
  HGB, D21: Above | 4 | 3 | 3 | 2
  LYM, PRE: number analyzed (Participants) | 37 | 37 | 28 | 28
  LYM, PRE: Unknown | 2 | 6 | 4 | 0
  LYM, PRE: Below | 0 | 0 | 1 | 0
  LYM, PRE: Within | 27 | 23 | 17 | 22
  LYM, PRE: Above | 8 | 8 | 6 | 6
  LYM, D7: Unknown | 5 | 4 | 4 | 3
  LYM, D7: Below | 1 | 2 | 0 | 0
  LYM, D7: Within | 38 | 28 | 33 | 44
  LYM, D7: Above | 22 | 26 | 23 | 14
  LYM, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  LYM, D21: Unknown | 1 | 3 | 6 | 0
  LYM, D21: Below | 0 | 1 | 0 | 1
  LYM, D21: Within | 43 | 27 | 35 | 38
  LYM, D21: Above | 21 | 26 | 17 | 22
  MON, PRE: number analyzed (Participants) | 37 | 37 | 28 | 28
  MON, PRE: Unknown | 2 | 6 | 4 | 0
  MON, PRE: Below | 4 | 5 | 3 | 5
  MON, PRE: Within | 31 | 26 | 21 | 22
  MON, PRE: Above | 0 | 0 | 0 | 1
  MON, D7: Unknown | 5 | 4 | 4 | 3
  MON, D7: Below | 13 | 10 | 11 | 7
  MON, D7: Within | 48 | 46 | 44 | 51
  MON, D7: Above | 0 | 0 | 1 | 0
  MON, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  MON, D21: Unknown | 1 | 3 | 6 | 0
  MON, D21: Below | 19 | 8 | 10 | 13
  MON, D21: Within | 45 | 46 | 42 | 48
  MON, D21: Above | 0 | 0 | 0 | 0
  NEU, PRE: number analyzed (Participants) | 37 | 37 | 28 | 28
  NEU, PRE: Unknown | 2 | 6 | 4 | 0
  NEU, PRE: Below | 3 | 2 | 0 | 3
  NEU, PRE: Within | 31 | 27 | 21 | 25
  NEU, PRE: Above | 1 | 2 | 3 | 0
  NEU, D7: Unknown | 5 | 4 | 4 | 3
  NEU, D7: Below | 10 | 3 | 2 | 6
  NEU, D7: Within | 50 | 52 | 54 | 50
  NEU, D7: Above | 1 | 1 | 0 | 2
  NEU, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  NEU, D21: Unknown | 1 | 3 | 6 | 0
  NEU, D21: Below | 1 | 3 | 3 | 2
  NEU, D21: Within | 62 | 51 | 49 | 59
  NEU, D21: Above | 1 | 0 | 0 | 0
  PLC, PRE: number analyzed (Participants) | 37 | 37 | 28 | 28
  PLC, PRE: Unknown | 2 | 7 | 5 | 1
  PLC, PRE: Below | 0 | 0 | 0 | 0
  PLC, PRE: Within | 33 | 26 | 20 | 27
  PLC, PRE: Above | 2 | 4 | 3 | 0
  PLC, D7: Unknown | 6 | 3 | 4 | 3
  PLC, D7: Below | 0 | 0 | 1 | 0
  PLC, D7: Within | 51 | 49 | 50 | 51
  PLC, D7: Above | 9 | 8 | 5 | 7
  PLC, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  PLC, D21: Unknown | 2 | 4 | 6 | 0
  PLC, D21: Below | 0 | 1 | 0 | 0
  PLC, D21: Within | 57 | 43 | 51 | 57
  PLC, D21: Above | 6 | 9 | 1 | 4
  RBC, PRE: number analyzed (Participants) | 37 | 37 | 28 | 28
  RBC, PRE: Unknown | 2 | 6 | 4 | 0
  RBC, PRE: Below | 0 | 1 | 0 | 2
  RBC, PRE: Within | 34 | 29 | 23 | 25
  RBC, PRE: Above | 1 | 1 | 1 | 1
  RBC, D7: Unknown | 5 | 4 | 4 | 3
  RBC, D7: Below | 2 | 3 | 1 | 1
  RBC, D7: Within | 56 | 52 | 54 | 54
  RBC, D7: Above | 3 | 1 | 1 | 3
  RBC, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  RBC, D21: Unknown | 1 | 3 | 6 | 0
  RBC, D21: Below | 1 | 3 | 2 | 1
  RBC, D21: Within | 62 | 51 | 48 | 57
  RBC, D21: Above | 1 | 0 | 2 | 3
  WBC, PRE: number analyzed (Participants) | 37 | 37 | 28 | 28
  WBC, PRE: Unknown | 2 | 6 | 4 | 0
  WBC, PRE: Below | 1 | 0 | 0 | 2
  WBC, PRE: Within | 33 | 30 | 22 | 26
  WBC, PRE: Above | 1 | 1 | 2 | 0
  WBC, D7: Unknown | 5 | 4 | 4 | 3
  WBC, D7: Below | 6 | 2 | 1 | 1
  WBC, D7: Within | 54 | 53 | 55 | 56
  WBC, D7: Above | 1 | 1 | 0 | 1
  WBC, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  WBC, D21: Unknown | 1 | 3 | 6 | 0
  WBC, D21: Below | 2 | 1 | 0 | 1
  WBC, D21: Within | 61 | 53 | 52 | 60
  WBC, D21: Above | 1 | 0 | 0 | 0

52. Secondary Outcome: Number of Subjects With Biochemical Laboratory Abnormalities - Preliminary Analysis
Description: Biochemical parameters assessed for lab abnormalities were alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin [BLR], bilirubin conjugated/direct [BCD], creatinine [CRE] and blood urea nitrogen [BUN]. Biochemical laboratory values were unknown, below, within or above the laboratory reference range defined for the specified time point and laboratory parameter.
Time Frame: At Day 0 (PRE), at Day 7 and at Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 66 | 60 | 60 | 61
Participants
  ALT, PRE: number analyzed (Participants) | 37 | 37 | 29 | 28
  ALT, PRE: Unkown | 0 | 2 | 2 | 0
  ALT, PRE: Below | 0 | 0 | 0 | 0
  ALT, PRE: Within | 37 | 35 | 27 | 28
  ALT, PRE: Above | 0 | 0 | 0 | 0
  ALT, D7: Unkown | 1 | 1 | 0 | 1
  ALT, D7: Below | 0 | 0 | 0 | 0
  ALT, D7: Within | 64 | 59 | 59 | 59
  ALT, D7: Above | 1 | 0 | 1 | 1
  ALT, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  ALT, D21: Unkown | 2 | 0 | 4 | 0
  ALT, D21: Below | 0 | 0 | 0 | 0
  ALT, D21: Within | 63 | 57 | 54 | 61
  ALT, D21: Above | 0 | 0 | 0 | 0
  AST, PRE: number analyzed (Participants) | 37 | 37 | 29 | 28
  AST, PRE: Unkown | 3 | 5 | 3 | 0
  AST, PRE: Below | 0 | 0 | 0 | 0
  AST, PRE: Within | 34 | 32 | 26 | 28
  AST, PRE: Above | 0 | 0 | 0 | 0
  AST, D7: Unkown | 1 | 3 | 0 | 1
  AST, D7: Below | 0 | 0 | 0 | 0
  AST, D7: Within | 63 | 57 | 57 | 58
  AST, D7: Above | 2 | 0 | 3 | 2
  AST, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  AST, D21: Unkown | 4 | 0 | 4 | 1
  AST, D21: Below | 0 | 0 | 0 | 0
  AST, D21: Within | 61 | 56 | 52 | 60
  AST, D21: Above | 0 | 1 | 2 | 0
  BLR, PRE: number analyzed (Participants) | 37 | 37 | 29 | 28
  BLR, PRE: Unkown | 0 | 2 | 2 | 0
  BLR, PRE: Below | 0 | 0 | 0 | 0
  BLR, PRE: Within | 37 | 35 | 27 | 28
  BLR, PRE: Above | 0 | 0 | 0 | 0
  BLR, D7: Unkown | 1 | 1 | 0 | 1
  BLR, D7: Below | 0 | 0 | 0 | 0
  BLR, D7: Within | 65 | 59 | 60 | 60
  BLR, D7: Above | 0 | 0 | 0 | 0
  BLR, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  BLR, D21: Unkown | 2 | 0 | 4 | 0
  BLR, D21: Below | 0 | 0 | 0 | 0
  BLR, D21: Within | 63 | 57 | 54 | 61
  BLR, D21: Above | 0 | 0 | 0 | 0
  BCD, PRE: number analyzed (Participants) | 37 | 37 | 29 | 28
  BCD, PRE: Unkown | 0 | 2 | 2 | 0
  BCD, PRE: Below | 0 | 0 | 0 | 0
  BCD, PRE: Within | 37 | 35 | 27 | 28
  BCD, PRE: Above | 0 | 0 | 0 | 0
  BCD, D7: Unkown | 1 | 1 | 0 | 1
  BCD, D7: Below | 0 | 0 | 0 | 0
  BCD, D7: Within | 65 | 59 | 60 | 60
  BCD, D7: Above | 0 | 0 | 0 | 0
  BCD, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  BCD, D21: Unkown | 2 | 0 | 4 | 0
  BCD, D21: Below | 0 | 0 | 0 | 0
  BCD, D21: Within | 63 | 57 | 54 | 61
  BCD, D21: Above | 0 | 0 | 0 | 0
  CRE, PRE: number analyzed (Participants) | 37 | 37 | 29 | 28
  CRE, PRE: Unkown | 0 | 2 | 2 | 0
  CRE, PRE: Below | 13 | 15 | 10 | 7
  CRE, PRE: Within | 24 | 20 | 17 | 21
  CRE, PRE: Above | 0 | 0 | 0 | 0
  CRE, D7: Unkown | 1 | 1 | 0 | 1
  CRE, D7: Below | 18 | 23 | 19 | 17
  CRE, D7: Within | 47 | 36 | 41 | 43
  CRE, D7: Above | 0 | 0 | 0 | 0
  CRE, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  CRE, D21: Unkown | 2 | 0 | 4 | 0
  CRE, D21: Below | 22 | 23 | 15 | 17
  CRE, D21: Within | 41 | 34 | 39 | 44
  CRE, D21: Above | 0 | 0 | 0 | 0
  BUN, PRE: number analyzed (Participants) | 37 | 37 | 29 | 28
  BUN, PRE: Unkown | 0 | 2 | 2 | 0
  BUN, PRE: Below | 1 | 0 | 0 | 0
  BUN, PRE: Within | 35 | 33 | 23 | 25
  BUN, PRE: Above | 1 | 2 | 4 | 3
  BUN, D7: Unkown | 1 | 1 | 0 | 1
  BUN, D7: Below | 0 | 0 | 0 | 1
  BUN, D7: Within | 62 | 55 | 51 | 51
  BUN, D7: Above | 3 | 4 | 9 | 8
  BUN, D21: number analyzed (Participants) | 65 | 57 | 58 | 61
  BUN, D21: Unkown | 2 | 0 | 4 | 0
  BUN, D21: Below | 0 | 0 | 0 | 0
  BUN, D21: Within | 59 | 54 | 48 | 52
  BUN, D21: Above | 4 | 3 | 6 | 9

53. Secondary Outcome: Number of Subjects With Haematological Laboratory Abnormalities - First Analysis
Description: as for outcome 51
Time Frame: At Day 0 (PRE), at Day 7, at Day 21 and at Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 66 | 63 | 63 | 63
Participants
  BAS, PRE: Unknown | 1 | 3 | 7 | 2
  BAS, PRE: Below | 0 | 0 | 0 | 0
  BAS, PRE: Within | 65 | 60 | 56 | 61
  BAS, PRE: Above | 0 | 0 | 0 | 0
  BAS, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  BAS, D7: Unknown | 5 | 4 | 4 | 3
  BAS, D7: Below | 0 | 0 | 0 | 0
  BAS, D7: Within | 61 | 56 | 56 | 58
  BAS, D7: Above | 0 | 0 | 0 | 0
  BAS, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  BAS, D21: Unknown | 1 | 3 | 6 | 0
  BAS, D21: Below | 0 | 0 | 0 | 0
  BAS, D21: Within | 64 | 54 | 53 | 61
  BAS, D21: Above | 0 | 0 | 0 | 0
  BAS, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  BAS, D42: Unknown | 3 | 2 | 1 | 1
  BAS, D42: Below | 0 | 0 | 0 | 0
  BAS, D42: Within | 55 | 54 | 59 | 57
  BAS, D42: Above | 0 | 0 | 0 | 0
  EOS, PRE: Unknown | 4 | 2 | 6 | 1
  EOS, PRE: Below | 12 | 5 | 7 | 6
  EOS, PRE: Within | 46 | 53 | 45 | 51
  EOS, PRE: Above | 4 | 3 | 5 | 5
  EOS, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  EOS, D7: Unknown | 5 | 4 | 4 | 3
  EOS, D7: Below | 7 | 8 | 8 | 6
  EOS, D7: Within | 50 | 42 | 46 | 45
  EOS, D7: Above | 4 | 6 | 2 | 7
  EOS, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  EOS, D21: Unknown | 1 | 3 | 6 | 0
  EOS, D21: Below | 5 | 6 | 5 | 7
  EOS, D21: Within | 54 | 42 | 47 | 51
  EOS, D21: Above | 5 | 6 | 1 | 3
  EOS, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  EOS, D42: Unknown | 3 | 2 | 1 | 1
  EOS, D42: Below | 4 | 3 | 5 | 3
  EOS, D42: Within | 42 | 46 | 50 | 47
  EOS, D42: Above | 9 | 5 | 4 | 7
  HCT, PRE: Unknown | 5 | 5 | 6 | 2
  HCT, PRE: Below | 5 | 8 | 4 | 5
  HCT, PRE: Within | 53 | 44 | 48 | 52
  HCT, PRE: Above | 3 | 6 | 5 | 4
  HCT, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  HCT, D7: Unknown | 5 | 4 | 4 | 3
  HCT, D7: Below | 6 | 7 | 4 | 6
  HCT, D7: Within | 52 | 47 | 48 | 49
  HCT, D7: Above | 3 | 2 | 4 | 3
  HCT, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  HCT, D21: Unknown | 1 | 3 | 6 | 0
  HCT, D21: Below | 7 | 10 | 7 | 7
  HCT, D21: Within | 54 | 41 | 43 | 53
  HCT, D21: Above | 3 | 3 | 3 | 1
  HCT, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  HCT, D42: Unknown | 3 | 2 | 1 | 1
  HCT, D42: Below | 9 | 12 | 5 | 10
  HCT, D42: Within | 45 | 41 | 48 | 46
  HCT, D42: Above | 1 | 1 | 6 | 1
  HGB, PRE: Unknown | 3 | 6 | 4 | 2
  HGB, PRE: Below | 1 | 5 | 3 | 3
  HGB, PRE: Within | 58 | 45 | 52 | 55
  HGB, PRE: Above | 4 | 7 | 4 | 3
  HGB, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  HGB, D7: Unknown | 5 | 3 | 4 | 3
  HGB, D7: Below | 4 | 5 | 1 | 2
  HGB, D7: Within | 55 | 50 | 51 | 52
  HGB, D7: Above | 2 | 2 | 4 | 4
  HGB, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  HGB, D21: Unknown | 1 | 3 | 6 | 0
  HGB, D21: Below | 5 | 3 | 3 | 3
  HGB, D21: Within | 55 | 48 | 47 | 56
  HGB, D21: Above | 4 | 3 | 3 | 2
  HGB, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  HGB, D42: Unknown | 3 | 2 | 1 | 1
  HGB, D42: Below | 2 | 8 | 4 | 4
  HGB, D42: Within | 49 | 43 | 49 | 50
  HGB, D42: Above | 4 | 3 | 6 | 3
  LYM, PRE: Unknown | 2 | 4 | 6 | 2
  LYM, PRE: Below | 0 | 0 | 1 | 0
  LYM, PRE: Within | 46 | 38 | 35 | 43
  LYM, PRE: Above | 18 | 21 | 21 | 18
  LYM, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  LYM, D7: Unknown | 5 | 4 | 4 | 3
  LYM, D7: Below | 1 | 2 | 0 | 0
  LYM, D7: Within | 38 | 28 | 33 | 44
  LYM, D7: Above | 22 | 26 | 23 | 14
  LYM, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  LYM, D21: Unknown | 1 | 3 | 6 | 0
  LYM, D21: Below | 0 | 1 | 0 | 1
  LYM, D21: Within | 43 | 27 | 36 | 38
  LYM, D21: Above | 21 | 26 | 17 | 22
  LYM, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  LYM, D42: Unknown | 3 | 2 | 1 | 1
  LYM, D42: Below | 1 | 1 | 0 | 0
  LYM, D42: Within | 36 | 31 | 36 | 40
  LYM, D42: Above | 18 | 22 | 23 | 17
  MON, PRE: Unknown | 4 | 5 | 6 | 1
  MON, PRE: Below | 10 | 10 | 4 | 15
  MON, PRE: Within | 52 | 48 | 53 | 46
  MON, PRE: Above | 0 | 0 | 0 | 1
  MON, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  MON, D7: Unknown | 5 | 4 | 4 | 3
  MON, D7: Below | 13 | 10 | 11 | 7
  MON, D7: Within | 48 | 46 | 44 | 51
  MON, D7: Above | 0 | 0 | 1 | 0
  MON, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  MON, D21: Unknown | 1 | 3 | 6 | 0
  MON, D21: Below | 19 | 8 | 10 | 13
  MON, D21: Within | 45 | 46 | 43 | 48
  MON, D21: Above | 0 | 0 | 0 | 0
  MON, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  MON, D42: Unknown | 3 | 2 | 1 | 1
  MON, D42: Below | 13 | 17 | 21 | 16
  MON, D42: Within | 41 | 37 | 38 | 41
  MON, D42: Above | 1 | 0 | 0 | 0
  NEU, PRE: Unknown | 5 | 4 | 4 | 1
  NEU, PRE: Below | 5 | 6 | 4 | 6
  NEU, PRE: Within | 54 | 52 | 51 | 56
  NEU, PRE: Above | 2 | 1 | 4 | 0
  NEU, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  NEU, D7: Unknown | 5 | 4 | 4 | 3
  NEU, D7: Below | 10 | 3 | 2 | 6
  NEU, D7: Within | 50 | 52 | 54 | 50
  NEU, D7: Above | 1 | 1 | 0 | 2
  NEU, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  NEU, D21: Unknown | 1 | 3 | 6 | 0
  NEU, D21: Below | 1 | 3 | 3 | 2
  NEU, D21: Within | 62 | 51 | 50 | 59
  NEU, D21: Above | 1 | 0 | 0 | 0
  NEU, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  NEU, D42: Unknown | 3 | 2 | 1 | 1
  NEU, D42: Below | 5 | 5 | 10 | 13
  NEU, D42: Within | 50 | 48 | 48 | 40
  NEU, D42: Above | 0 | 1 | 1 | 4
  PLC, PRE: Unknown | 4 | 8 | 8 | 3
  PLC, PRE: Below | 0 | 0 | 1 | 0
  PLC, PRE: Within | 51 | 49 | 48 | 56
  PLC, PRE: Above | 11 | 6 | 6 | 4
  PLC, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  PLC, D7: Unknown | 6 | 3 | 4 | 3
  PLC, D7: Below | 0 | 0 | 1 | 0
  PLC, D7: Within | 51 | 49 | 50 | 51
  PLC, D7: Above | 9 | 8 | 5 | 7
  PLC, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  PLC, D21: Unknown | 2 | 4 | 6 | 0
  PLC, D21: Below | 0 | 1 | 0 | 0
  PLC, D21: Within | 57 | 43 | 52 | 57
  PLC, D21: Above | 6 | 9 | 1 | 4
  PLC, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  PLC, D42: Unknown | 3 | 3 | 1 | 2
  PLC, D42: Below | 0 | 0 | 0 | 1
  PLC, D42: Within | 50 | 47 | 59 | 53
  PLC, D42: Above | 5 | 6 | 0 | 2
  RBC, PRE: Unknown | 4 | 4 | 5 | 2
  RBC, PRE: Below | 1 | 4 | 0 | 3
  RBC, PRE: Within | 59 | 54 | 56 | 55
  RBC, PRE: Above | 2 | 1 | 2 | 3
  RBC, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  RBC, D7: Unknown | 5 | 4 | 4 | 3
  RBC, D7: Below | 2 | 3 | 1 | 1
  RBC, D7: Within | 56 | 52 | 54 | 54
  RBC, D7: Above | 3 | 1 | 1 | 3
  RBC, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  RBC, D21: Unknown | 1 | 3 | 6 | 0
  RBC, D21: Below | 1 | 3 | 2 | 1
  RBC, D21: Within | 62 | 51 | 49 | 57
  RBC, D21: Above | 1 | 0 | 2 | 3
  RBC, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  RBC, D42: Unknown | 3 | 2 | 1 | 1
  RBC, D42: Below | 1 | 2 | 2 | 3
  RBC, D42: Within | 51 | 52 | 55 | 52
  RBC, D42: Above | 3 | 0 | 2 | 2
  WBC, PRE: Unknown | 6 | 5 | 6 | 2
  WBC, PRE: Below | 3 | 0 | 1 | 2
  WBC, PRE: Within | 55 | 57 | 54 | 59
  WBC, PRE: Above | 2 | 1 | 2 | 0
  WBC, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  WBC, D7: Unknown | 5 | 4 | 4 | 3
  WBC, D7: Below | 6 | 2 | 1 | 1
  WBC, D7: Within | 54 | 53 | 55 | 56
  WBC, D7: Above | 1 | 1 | 0 | 1
  WBC, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  WBC, D21: Unknown | 1 | 3 | 6 | 0
  WBC, D21: Below | 2 | 1 | 0 | 1
  WBC, D21: Within | 61 | 53 | 53 | 60
  WBC, D21: Above | 1 | 0 | 0 | 0
  WBC, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  WBC, D42: Unknown | 3 | 2 | 1 | 1
  WBC, D42: Below | 3 | 3 | 2 | 5
  WBC, D42: Within | 52 | 51 | 56 | 50
  WBC, D42: Above | 0 | 0 | 1 | 2

54. Secondary Outcome: Number of Subjects With Biochemical Laboratory Abnormalities - First Analysis
Description: as for outcome 52
Time Frame: At Day 0 (PRE), at Day 7, at Day 21 and at Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 66 | 63 | 63 | 63
Participants
  ALT, PRE: Unknown | 2 | 2 | 3 | 0
  ALT, PRE: Below | 0 | 0 | 0 | 0
  ALT, PRE: Within | 64 | 61 | 59 | 63
  ALT, PRE: Above | 0 | 0 | 1 | 0
  ALT, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  ALT, D7: Unknown | 1 | 1 | 0 | 1
  ALT, D7: Below | 0 | 0 | 0 | 0
  ALT, D7: Within | 64 | 59 | 59 | 59
  ALT, D7: Above | 1 | 0 | 1 | 1
  ALT, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  ALT, D21: Unknown | 2 | 0 | 4 | 0
  ALT, D21: Below | 0 | 0 | 0 | 0
  ALT, D21: Within | 63 | 57 | 55 | 61
  ALT, D21: Above | 0 | 0 | 0 | 0
  ALT, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  ALT, D42: Unknown | 3 | 2 | 0 | 1
  ALT, D42: Below | 0 | 0 | 0 | 0
  ALT, D42: Within | 55 | 53 | 59 | 56
  ALT, D42: Above | 0 | 1 | 1 | 1
  AST, PRE: Unknown | 5 | 6 | 3 | 0
  AST, PRE: Below | 0 | 0 | 0 | 0
  AST, PRE: Within | 61 | 57 | 59 | 63
  AST, PRE: Above | 0 | 0 | 1 | 0
  AST, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  AST, D7: Unknown | 1 | 3 | 0 | 1
  AST, D7: Below | 0 | 0 | 0 | 0
  AST, D7: Within | 63 | 57 | 57 | 58
  AST, D7: Above | 2 | 0 | 3 | 2
  AST, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  AST, D21: Unknown | 4 | 0 | 4 | 1
  AST, D21: Below | 0 | 0 | 0 | 0
  AST, D21: Within | 61 | 56 | 53 | 60
  AST, D21: Above | 0 | 1 | 2 | 0
  AST, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  AST, D42: Unknown | 4 | 2 | 0 | 1
  AST, D42: Below | 0 | 0 | 0 | 0
  AST, D42: Within | 54 | 53 | 57 | 57
  AST, D42: Above | 0 | 1 | 3 | 0
  BLR, PRE: Unknown | 2 | 1 | 3 | 0
  BLR, PRE: Below | 0 | 0 | 0 | 0
  BLR, PRE: Within | 64 | 62 | 60 | 63
  BLR, PRE: Above | 0 | 0 | 0 | 0
  BLR, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  BLR, D7: Unknown | 1 | 1 | 0 | 1
  BLR, D7: Below | 0 | 0 | 0 | 0
  BLR, D7: Within | 65 | 59 | 60 | 60
  BLR, D7: Above | 0 | 0 | 0 | 0
  BLR, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  BLR, D21: Unknown | 2 | 0 | 4 | 0
  BLR, D21: Below | 0 | 0 | 0 | 0
  BLR, D21: Within | 63 | 57 | 55 | 61
  BLR, D21: Above | 0 | 0 | 0 | 0
  BLR, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  BLR, D42: Unknown | 3 | 2 | 0 | 1
  BLR, D42: Below | 0 | 0 | 0 | 0
  BLR, D42: Within | 55 | 53 | 60 | 57
  BLR, D42: Above | 0 | 1 | 0 | 0
  BCD, PRE: Unknown | 2 | 2 | 3 | 0
  BCD, PRE: Below | 0 | 0 | 0 | 0
  BCD, PRE: Within | 64 | 61 | 60 | 63
  BCD, PRE: Above | 0 | 0 | 0 | 0
  BCD, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  BCD, D7: Unknown | 1 | 1 | 0 | 1
  BCD, D7: Below | 0 | 0 | 0 | 0
  BCD, D7: Within | 65 | 59 | 60 | 60
  BCD, D7: Above | 0 | 0 | 0 | 0
  BCD, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  BCD, D21: Unknown | 2 | 0 | 4 | 0
  BCD, D21: Below | 0 | 0 | 0 | 0
  BCD, D21: Within | 63 | 57 | 55 | 61
  BCD, D21: Above | 0 | 0 | 0 | 0
  BCD, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  BCD, D42: Unknown | 3 | 2 | 0 | 1
  BCD, D42: Below | 0 | 0 | 0 | 0
  BCD, D42: Within | 55 | 54 | 60 | 57
  BCD, D42: Above | 0 | 0 | 0 | 0
  CRE, PRE: Unknown | 2 | 2 | 3 | 0
  CRE, PRE: Below | 19 | 22 | 17 | 15
  CRE, PRE: Within | 45 | 39 | 43 | 48
  CRE, PRE: Above | 0 | 0 | 0 | 0
  CRE, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  CRE, D7: Unknown | 1 | 1 | 0 | 1
  CRE, D7: Below | 18 | 23 | 19 | 17
  CRE, D7: Within | 47 | 36 | 41 | 43
  CRE, D7: Above | 0 | 0 | 0 | 0
  CRE, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  CRE, D21: Unknown | 2 | 0 | 4 | 0
  CRE, D21: Below | 22 | 23 | 15 | 17
  CRE, D21: Within | 41 | 34 | 40 | 44
  CRE, D21: Above | 0 | 0 | 0 | 0
  CRE, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  CRE, D42: Unknown | 3 | 2 | 0 | 1
  CRE, D42: Below | 18 | 20 | 16 | 13
  CRE, D42: Within | 37 | 34 | 44 | 44
  CRE, D42: Above | 0 | 0 | 0 | 0
  BUN, PRE: Unknown | 2 | 2 | 3 | 0
  BUN, PRE: Below | 2 | 0 | 0 | 0
  BUN, PRE: Within | 58 | 55 | 55 | 58
  BUN, PRE: Above | 4 | 6 | 5 | 5
  BUN, D7: number analyzed (Participants) | 66 | 60 | 60 | 61
  BUN, D7: Unknown | 1 | 1 | 0 | 1
  BUN, D7: Below | 0 | 0 | 0 | 1
  BUN, D7: Within | 62 | 55 | 51 | 51
  BUN, D7: Above | 3 | 4 | 9 | 8
  BUN, D21: number analyzed (Participants) | 65 | 57 | 59 | 61
  BUN, D21: Unknown | 2 | 0 | 4 | 0
  BUN, D21: Below | 0 | 0 | 0 | 0
  BUN, D21: Within | 59 | 54 | 49 | 52
  BUN, D21: Above | 4 | 3 | 6 | 9
  BUN, D42: number analyzed (Participants) | 58 | 56 | 60 | 58
  BUN, D42: Unknown | 3 | 2 | 0 | 1
  BUN, D42: Below | 1 | 0 | 0 | 0
  BUN, D42: Within | 49 | 49 | 54 | 50
  BUN, D42: Above | 5 | 5 | 6 | 7

55. Secondary Outcome: Number of Subjects With Haematological Laboratory Abnormalities - Second Analysis
Description: Among haematological parameters assessed were basophils [BAS], eosinophils [EOS], hematocrit [HCT], hemoglobin level [HGB], lymphocytes [LYM], monocytes [MON], neutrophils [NEU], platelet count [PLC], red blood cells [RBC] and white blood cells [WBC], Haematological laboratory values were unknown, below, within or above the laboratory reference range defined for the specified time point and laboratory parameter.
Time Frame: At Day 0 (PRE), at Day 7 and at Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 66 | 126 | 63 | 63
Participants
  BAS, PRE: Unknown | 1 | 5 | 3 | 1
  BAS, PRE: Below | 0 | 0 | 0 | 0
  BAS, PRE: Within | 65 | 121 | 60 | 62
  BAS, PRE: Above | 0 | 0 | 0 | 0
  BAS, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  BAS, D7: Unknown | 5 | 5 | 4 | 3
  BAS, D7: Below | 0 | 0 | 0 | 0
  BAS, D7: Within | 61 | 115 | 56 | 58
  BAS, D7: Above | 0 | 0 | 0 | 0
  BAS, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  BAS, D21: Unknown | 1 | 4 | 6 | 0
  BAS, D21: Below | 0 | 0 | 0 | 0
  BAS, D21: Within | 64 | 112 | 53 | 61
  BAS, D21: Above | 0 | 0 | 0 | 0
  BAS, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  BAS, D42: Unknown | 3 | 5 | 1 | 1
  BAS, D42: Below | 0 | 0 | 0 | 0
  BAS, D42: Within | 55 | 109 | 59 | 57
  BAS, D42: Above | 0 | 0 | 0 | 0
  EOS, PRE: Unknown | 1 | 5 | 3 | 1
  EOS, PRE: Below | 12 | 11 | 7 | 6
  EOS, PRE: Within | 49 | 100 | 48 | 51
  EOS, PRE: Above | 4 | 10 | 5 | 5
  EOS, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  EOS, D7: Unknown | 5 | 5 | 4 | 3
  EOS, D7: Below | 7 | 20 | 8 | 6
  EOS, D7: Within | 50 | 84 | 46 | 45
  EOS, D7: Above | 4 | 11 | 2 | 7
  EOS, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  EOS, D21: Unknown | 1 | 4 | 6 | 0
  EOS, D21: Below | 5 | 14 | 5 | 7
  EOS, D21: Within | 54 | 90 | 47 | 51
  EOS, D21: Above | 5 | 8 | 1 | 3
  EOS, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  EOS, D42: Unknown | 3 | 5 | 1 | 1
  EOS, D42: Below | 4 | 8 | 5 | 3
  EOS, D42: Within | 42 | 94 | 50 | 47
  EOS, D42: Above | 9 | 7 | 4 | 7
  HCT, PRE: Unknown | 1 | 6 | 3 | 1
  HCT, PRE: Below | 5 | 22 | 5 | 6
  HCT, PRE: Within | 56 | 90 | 50 | 52
  HCT, PRE: Above | 4 | 8 | 5 | 4
  HCT, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  HCT, D7: Unknown | 5 | 5 | 4 | 3
  HCT, D7: Below | 6 | 26 | 4 | 6
  HCT, D7: Within | 52 | 82 | 48 | 49
  HCT, D7: Above | 3 | 7 | 4 | 3
  HCT, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  HCT, D21: Unknown | 1 | 4 | 6 | 0
  HCT, D21: Below | 7 | 32 | 7 | 7
  HCT, D21: Within | 54 | 77 | 43 | 53
  HCT, D21: Above | 3 | 3 | 3 | 1
  HCT, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  HCT, D42: Unknown | 3 | 6 | 1 | 1
  HCT, D42: Below | 9 | 24 | 5 | 10
  HCT, D42: Within | 45 | 80 | 48 | 46
  HCT, D42: Above | 1 | 4 | 6 | 1
  HGB, PRE: Unknown | 1 | 5 | 3 | 1
  HGB, PRE: Below | 1 | 15 | 3 | 4
  HGB, PRE: Within | 59 | 96 | 53 | 55
  HGB, PRE: Above | 5 | 10 | 4 | 3
  HGB, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  HGB, D7: Unknown | 5 | 4 | 4 | 3
  HGB, D7: Below | 4 | 9 | 1 | 2
  HGB, D7: Within | 55 | 98 | 51 | 52
  HGB, D7: Above | 2 | 9 | 4 | 4
  HGB, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  HGB, D21: Unknown | 1 | 4 | 6 | 0
  HGB, D21: Below | 5 | 10 | 3 | 3
  HGB, D21: Within | 55 | 97 | 47 | 56
  HGB, D21: Above | 4 | 5 | 3 | 2
  HGB, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  HGB, D42: Unknown | 3 | 5 | 1 | 1
  HGB, D42: Below | 2 | 13 | 4 | 4
  HGB, D42: Within | 49 | 90 | 49 | 50
  HGB, D42: Above | 4 | 6 | 6 | 3
  LYM, PRE: Unknown | 1 | 5 | 3 | 1
  LYM, PRE: Below | 0 | 1 | 1 | 0
  LYM, PRE: Within | 47 | 83 | 37 | 44
  LYM, PRE: Above | 18 | 37 | 22 | 18
  LYM, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  LYM, D7: Unknown | 5 | 5 | 4 | 3
  LYM, D7: Below | 1 | 3 | 0 | 0
  LYM, D7: Within | 38 | 73 | 33 | 44
  LYM, D7: Above | 22 | 39 | 23 | 14
  LYM, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  LYM, D21: Unknown | 1 | 4 | 6 | 0
  LYM, D21: Below | 0 | 2 | 0 | 1
  LYM, D21: Within | 43 | 72 | 36 | 38
  LYM, D21: Above | 21 | 38 | 17 | 22
  LYM, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  LYM, D42: Unknown | 3 | 5 | 1 | 1
  LYM, D42: Below | 1 | 3 | 0 | 0
  LYM, D42: Within | 36 | 75 | 36 | 40
  LYM, D42: Above | 18 | 31 | 23 | 17
  MON, PRE: Unknown | 1 | 5 | 3 | 1
  MON, PRE: Below | 12 | 26 | 7 | 15
  MON, PRE: Within | 53 | 95 | 53 | 46
  MON, PRE: Above | 0 | 0 | 0 | 1
  MON, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  MON, D7: Unknown | 5 | 5 | 4 | 3
  MON, D7: Below | 13 | 19 | 11 | 7
  MON, D7: Within | 48 | 96 | 44 | 51
  MON, D7: Above | 0 | 0 | 1 | 0
  MON, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  MON, D21: Unknown | 1 | 4 | 6 | 0
  MON, D21: Below | 19 | 18 | 10 | 13
  MON, D21: Within | 45 | 94 | 43 | 48
  MON, D21: Above | 0 | 0 | 0 | 0
  MON, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  MON, D42: Unknown | 3 | 5 | 1 | 1
  MON, D42: Below | 13 | 22 | 21 | 16
  MON, D42: Within | 41 | 87 | 38 | 41
  MON, D42: Above | 1 | 0 | 0 | 0
  NEU, PRE: Unknown | 1 | 5 | 3 | 1
  NEU, PRE: Below | 6 | 9 | 4 | 6
  NEU, PRE: Within | 57 | 109 | 52 | 56
  NEU, PRE: Above | 2 | 3 | 4 | 0
  NEU, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  NEU, D7: Unknown | 5 | 5 | 4 | 3
  NEU, D7: Below | 10 | 4 | 2 | 6
  NEU, D7: Within | 50 | 109 | 54 | 50
  NEU, D7: Above | 1 | 2 | 0 | 2
  NEU, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  NEU, D21: Unknown | 1 | 4 | 6 | 0
  NEU, D21: Below | 1 | 10 | 3 | 2
  NEU, D21: Within | 62 | 100 | 50 | 59
  NEU, D21: Above | 1 | 2 | 0 | 0
  NEU, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  NEU, D42: Unknown | 3 | 5 | 1 | 1
  NEU, D42: Below | 5 | 12 | 10 | 13
  NEU, D42: Within | 50 | 96 | 48 | 40
  NEU, D42: Above | 0 | 1 | 1 | 4
  PLC, PRE: Unknown | 1 | 6 | 5 | 2
  PLC, PRE: Below | 0 | 1 | 1 | 0
  PLC, PRE: Within | 54 | 107 | 51 | 57
  PLC, PRE: Above | 11 | 12 | 6 | 4
  PLC, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  PLC, D7: Unknown | 6 | 5 | 4 | 3
  PLC, D7: Below | 0 | 0 | 1 | 0
  PLC, D7: Within | 51 | 95 | 50 | 51
  PLC, D7: Above | 9 | 20 | 5 | 7
  PLC, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  PLC, D21: Unknown | 2 | 7 | 6 | 0
  PLC, D21: Below | 0 | 2 | 0 | 0
  PLC, D21: Within | 57 | 89 | 52 | 57
  PLC, D21: Above | 6 | 18 | 1 | 4
  PLC, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  PLC, D42: Unknown | 3 | 6 | 1 | 2
  PLC, D42: Below | 0 | 0 | 0 | 1
  PLC, D42: Within | 50 | 93 | 59 | 53
  PLC, D42: Above | 5 | 15 | 0 | 2
  RBC, PRE: Unknown | 1 | 6 | 3 | 1
  RBC, PRE: Below | 1 | 6 | 0 | 3
  RBC, PRE: Within | 62 | 113 | 58 | 56
  RBC, PRE: Above | 2 | 1 | 2 | 3
  RBC, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  RBC, D7: Unknown | 5 | 5 | 4 | 3
  RBC, D7: Below | 2 | 4 | 1 | 1
  RBC, D7: Within | 56 | 110 | 54 | 54
  RBC, D7: Above | 3 | 1 | 1 | 3
  RBC, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  RBC, D21: Unknown | 1 | 4 | 6 | 0
  RBC, D21: Below | 1 | 5 | 2 | 1
  RBC, D21: Within | 62 | 107 | 49 | 57
  RBC, D21: Above | 1 | 0 | 2 | 3
  RBC, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  RBC, D42: Unknown | 3 | 6 | 1 | 1
  RBC, D42: Below | 1 | 4 | 2 | 3
  RBC, D42: Within | 51 | 103 | 55 | 52
  RBC, D42: Above | 3 | 1 | 2 | 2
  WBC, PRE: Unknown | 1 | 5 | 3 | 1
  WBC, PRE: Below | 4 | 0 | 1 | 2
  WBC, PRE: Within | 59 | 118 | 57 | 60
  WBC, PRE: Above | 2 | 3 | 2 | 0
  WBC, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  WBC, D7: Unknown | 5 | 5 | 4 | 3
  WBC, D7: Below | 6 | 3 | 1 | 1
  WBC, D7: Within | 54 | 110 | 55 | 56
  WBC, D7: Above | 1 | 2 | 0 | 1
  WBC, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  WBC, D21: Unknown | 1 | 4 | 6 | 0
  WBC, D21: Below | 2 | 4 | 0 | 1
  WBC, D21: Within | 61 | 107 | 53 | 60
  WBC, D21: Above | 1 | 1 | 0 | 0
  WBC, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  WBC, D42: Unknown | 3 | 5 | 1 | 1
  WBC, D42: Below | 3 | 7 | 2 | 5
  WBC, D42: Within | 52 | 102 | 56 | 50
  WBC, D42: Above | 0 | 0 | 1 | 2

56. Secondary Outcome: Number of Subjects With Biochemical Laboratory Abnormalities - Second Analysis
Description: as for outcome 52
Time Frame: At Day 0 (PRE), at Day 7, at Day 21 and at Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 66 | 126 | 63 | 63
Participants
  ALT, PRE: Unknown | 2 | 2 | 3 | 0
  ALT, PRE: Below | 0 | 0 | 0 | 0
  ALT, PRE: Within | 64 | 124 | 59 | 63
  ALT, PRE: Above | 0 | 0 | 1 | 0
  ALT, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  ALT, D7: Unknown | 1 | 2 | 0 | 1
  ALT, D7: Below | 0 | 0 | 0 | 0
  ALT, D7: Within | 64 | 118 | 59 | 59
  ALT, D7: Above | 1 | 0 | 1 | 1
  ALT, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  ALT, D21: Unknown | 2 | 0 | 4 | 0
  ALT, D21: Below | 0 | 0 | 0 | 0
  ALT, D21: Within | 63 | 115 | 55 | 61
  ALT, D21: Above | 0 | 1 | 0 | 0
  ALT, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  ALT, D42: Unknown | 3 | 3 | 0 | 1
  ALT, D42: Below | 0 | 0 | 0 | 0
  ALT, D42: Within | 55 | 110 | 59 | 56
  ALT, D42: Above | 0 | 1 | 1 | 1
  AST, PRE: Unknown | 4 | 4 | 3 | 0
  AST, PRE: Below | 0 | 0 | 0 | 0
  AST, PRE: Within | 62 | 117 | 59 | 63
  AST, PRE: Above | 0 | 5 | 1 | 0
  AST, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  AST, D7: Unknown | 1 | 4 | 0 | 1
  AST, D7: Below | 0 | 0 | 0 | 0
  AST, D7: Within | 63 | 113 | 57 | 58
  AST, D7: Above | 2 | 3 | 3 | 2
  AST, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  AST, D21: Unknown | 4 | 1 | 4 | 1
  AST, D21: Below | 0 | 0 | 0 | 0
  AST, D21: Within | 61 | 112 | 53 | 60
  AST, D21: Above | 0 | 3 | 2 | 0
  AST, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  AST, D42: Unknown | 4 | 3 | 0 | 1
  AST, D42: Below | 0 | 0 | 0 | 0
  AST, D42: Within | 54 | 105 | 57 | 57
  AST, D42: Above | 0 | 6 | 3 | 0
  BLR, PRE: Unknown | 2 | 2 | 3 | 0
  BLR, PRE: Below | 0 | 0 | 0 | 0
  BLR, PRE: Within | 64 | 124 | 60 | 63
  BLR, PRE: Above | 0 | 0 | 0 | 0
  BLR, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  BLR, D7: Unknown | 1 | 2 | 0 | 1
  BLR, D7: Below | 0 | 0 | 0 | 0
  BLR, D7: Within | 65 | 118 | 60 | 60
  BLR, D7: Above | 0 | 0 | 0 | 0
  BLR, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  BLR, D21: Unknown | 2 | 0 | 4 | 0
  BLR, D21: Below | 0 | 0 | 0 | 0
  BLR, D21: Within | 63 | 116 | 55 | 61
  BLR, D21: Above | 0 | 0 | 0 | 0
  BLR, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  BLR, D42: Unknown | 3 | 3 | 0 | 1
  BLR, D42: Below | 0 | 0 | 0 | 0
  BLR, D42: Within | 55 | 110 | 60 | 57
  BLR, D42: Above | 0 | 1 | 0 | 0
  BCD, PRE: Unknown | 2 | 2 | 3 | 0
  BCD, PRE: Below | 0 | 0 | 0 | 0
  BCD, PRE: Within | 64 | 124 | 60 | 63
  BCD, PRE: Above | 0 | 0 | 0 | 0
  BCD, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  BCD, D7: Unknown | 1 | 2 | 0 | 1
  BCD, D7: Below | 0 | 0 | 0 | 0
  BCD, D7: Within | 65 | 118 | 60 | 60
  BCD, D7: Above | 0 | 0 | 0 | 0
  BCD, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  BCD, D21: Unknown | 2 | 0 | 4 | 0
  BCD, D21: Below | 0 | 0 | 0 | 0
  BCD, D21: Within | 63 | 116 | 55 | 61
  BCD, D21: Above | 0 | 0 | 0 | 0
  BCD, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  BCD, D42: Unknown | 3 | 3 | 0 | 1
  BCD, D42: Below | 0 | 0 | 0 | 0
  BCD, D42: Within | 55 | 111 | 60 | 57
  BCD, D42: Above | 0 | 0 | 0 | 0
  CRE, PRE: Unknown | 2 | 2 | 3 | 0
  CRE, PRE: Below | 19 | 38 | 17 | 15
  CRE, PRE: Within | 45 | 86 | 43 | 48
  CRE, PRE: Above | 0 | 0 | 0 | 0
  CRE, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  CRE, D7: Unknown | 1 | 2 | 0 | 1
  CRE, D7: Below | 18 | 38 | 19 | 17
  CRE, D7: Within | 47 | 80 | 41 | 43
  CRE, D7: Above | 0 | 0 | 0 | 0
  CRE, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  CRE, D21: Unknown | 2 | 0 | 4 | 0
  CRE, D21: Below | 22 | 40 | 15 | 17
  CRE, D21: Within | 41 | 76 | 40 | 44
  CRE, D21: Above | 0 | 0 | 0 | 0
  CRE, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  CRE, D42: Unknown | 3 | 3 | 0 | 1
  CRE, D42: Below | 18 | 37 | 16 | 13
  CRE, D42: Within | 37 | 74 | 44 | 44
  CRE, D42: Above | 0 | 0 | 0 | 0
  BUN, PRE: Unknown | 2 | 2 | 3 | 0
  BUN, PRE: Below | 2 | 4 | 0 | 0
  BUN, PRE: Within | 58 | 110 | 56 | 58
  BUN, PRE: Above | 4 | 10 | 4 | 5
  BUN, D7: number analyzed (Participants) | 66 | 120 | 60 | 61
  BUN, D7: Unknown | 1 | 2 | 0 | 1
  BUN, D7: Below | 0 | 1 | 0 | 1
  BUN, D7: Within | 62 | 110 | 51 | 51
  BUN, D7: Above | 3 | 7 | 9 | 8
  BUN, D21: number analyzed (Participants) | 65 | 116 | 59 | 61
  BUN, D21: Unknown | 2 | 0 | 4 | 0
  BUN, D21: Below | 0 | 4 | 0 | 0
  BUN, D21: Within | 59 | 107 | 49 | 52
  BUN, D21: Above | 4 | 5 | 6 | 9
  BUN, D42: number analyzed (Participants) | 58 | 114 | 60 | 58
  BUN, D42: Unknown | 3 | 3 | 0 | 1
  BUN, D42: Below | 1 | 4 | 0 | 0
  BUN, D42: Within | 49 | 96 | 54 | 50
  BUN, D42: Above | 5 | 11 | 6 | 7

57. Secondary Outcome: Number of Subjects With Haematological Laboratory Abnormalities
Description: as for outcome 51
Time Frame: At Day 182
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 59 | 108 | 53 | 56
Participants
  BAS: Unknown | 5 | 8 | 2 | 3
  BAS: Below | 0 | 0 | 0 | 0
  BAS: Within | 54 | 100 | 51 | 53
  BAS: Above | 0 | 0 | 0 | 0
  EOS: Unknown | 5 | 8 | 2 | 3
  EOS: Below | 6 | 10 | 8 | 3
  EOS: Within | 43 | 83 | 39 | 47
  EOS: Above | 5 | 7 | 4 | 3
  HCT: Unknown | 5 | 9 | 3 | 3
  HCT: Below | 8 | 17 | 5 | 7
  HCT: Within | 43 | 70 | 42 | 43
  HCT: Above | 3 | 12 | 3 | 3
  HGB: Unknown | 5 | 8 | 2 | 3
  HGB: Below | 1 | 8 | 3 | 4
  HGB: Within | 50 | 79 | 44 | 45
  HGB: Above | 3 | 13 | 4 | 4
  LYM: Unknown | 5 | 8 | 2 | 3
  LYM: Below | 1 | 0 | 0 | 0
  LYM: Within | 40 | 72 | 37 | 41
  LYM: Above | 13 | 28 | 14 | 12
  MON: Unknown | 5 | 8 | 2 | 3
  MON: Below | 18 | 18 | 12 | 13
  MON: Within | 35 | 82 | 39 | 40
  MON: Above | 1 | 0 | 0 | 0
  NEU: Unknown | 5 | 8 | 2 | 3
  NEU: Below | 4 | 8 | 5 | 1
  NEU: Within | 48 | 92 | 43 | 51
  NEU: Above | 2 | 0 | 3 | 1
  PLC: Unknown | 6 | 9 | 2 | 3
  PLC: Below | 0 | 1 | 0 | 0
  PLC: Within | 48 | 92 | 51 | 52
  PLC: Above | 5 | 6 | 0 | 1
  RBC: Unknown | 5 | 9 | 3 | 3
  RBC: Below | 2 | 6 | 3 | 1
  RBC: Within | 51 | 91 | 47 | 51
  RBC: Above | 1 | 2 | 0 | 1
  WBC: Unknown | 5 | 8 | 2 | 3
  WBC: Below | 5 | 2 | 2 | 1
  WBC: Within | 49 | 98 | 47 | 51
  WBC: Above | 0 | 0 | 2 | 1

58. Secondary Outcome: Number of Subjects With Biochemical Laboratory Abnormalities
Description: as for outcome 52
Time Frame: At Day 182
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 59 | 108 | 53 | 56
Participants
  ALT: Unknown | 1 | 1 | 1 | 1
  ALT: Below | 0 | 0 | 0 | 0
  ALT: Within | 58 | 107 | 51 | 54
  ALT: Above | 0 | 0 | 1 | 1
  AST: Unknown | 1 | 1 | 1 | 2
  AST: Below | 0 | 0 | 0 | 0
  AST: Within | 57 | 106 | 50 | 53
  AST: Above | 1 | 1 | 2 | 1
  BLR: Unknown | 1 | 1 | 1 | 1
  BLR: Below | 0 | 0 | 0 | 0
  BLR: Within | 58 | 107 | 52 | 55
  BLR: Above | 0 | 0 | 0 | 0
  BCD: Unknown | 1 | 1 | 1 | 1
  BCD: Below | 0 | 0 | 0 | 0
  BCD: Within | 58 | 106 | 52 | 55
  BCD: Above | 0 | 1 | 0 | 0
  CRE: Unknown | 1 | 1 | 1 | 1
  CRE: Below | 18 | 35 | 16 | 18
  CRE: Within | 40 | 72 | 36 | 37
  CRE: Above | 0 | 0 | 0 | 0
  BUN: Unknown | 1 | 1 | 1 | 1
  BUN: Below | 3 | 2 | 1 | 0
  BUN: Within | 51 | 99 | 48 | 53
  BUN: Above | 4 | 6 | 3 | 2

59. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) - Preliminary Analysis
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 21 days (Days 0-20) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 64 | 64 | 63
Participants | 17 | 20 | 16 | 14

60. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) - First Analysis
Description: as for outcome 59
Time Frame: Within 42 days (Days 0-41) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 64 | 64 | 63
Participants | 33 | 35 | 25 | 23

61. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) - Second Analysis
Description: as for outcome 59
Time Frame: Within 41 days (Days 0-40) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 128 | 64 | 63
Participants | 34 | 65 | 24 | 23

62. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: as for outcome 59
Time Frame: Within 84 days (Days 0-83) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 128 | 64 | 63
Participants | 36 | 76 | 30 | 32

63. Secondary Outcome: Number of Subjects With Any Medically-attended Adverse Events (MAEs) - Preliminary Analysis
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination.
Time Frame: Within 21 days (Days 0-20) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 64 | 64 | 63
Participants | 7 | 5 | 3 | 4

64. Secondary Outcome: Number of Subjects With Any Medically-attended Adverse Events (MAEs) - First Analysis
Description: as for outcome 63
Time Frame: Within 41 days (Days 0-40) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 64 | 64 | 63
Participants | 18 | 14 | 8 | 9

65. Secondary Outcome: Number of Subjects With Any Medically-attended Adverse Events (MAEs) - Second Analysis
Description: as for outcome 63
Time Frame: Within 42 days (Days 0-41) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 128 | 64 | 63
Participants | 18 | 31 | 8 | 9

66. Secondary Outcome: Number of Subjects With Any Medically-attended Adverse Events (MAEs)
Description: as for outcome 63
Time Frame: Within 182 days (Days 0-181) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 128 | 64 | 63
Participants | 32 | 62 | 24 | 25

67. Secondary Outcome: Number of Subjects With Any Medically-attended Adverse Events (MAEs)
Description: as for outcome 63
Time Frame: Throughout the entire study period (Day 0 - Day 385)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 128 | 64 | 63
Participants | 39 | 87 | 39 | 34

68. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-mediated Diseases (pIMDs) - Preliminary Analysis
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: Within 21 days (Days 0-20) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 64 | 64 | 63
Participants | 0 | 0 | 0 | 0

69. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-mediated Diseases (pIMDs) - First Analysis
Description: as for outcome 68
Time Frame: Within 42 days (Days 0-41) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 64 | 64 | 63
Participants | 0 | 0 | 0 | 0

70. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-mediated Diseases (pIMDs) - Second Analysis
Description: as for outcome 68
Time Frame: Within 42 days (Days 0-41) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 128 | 64 | 63
Participants | 0 | 0 | 0 | 0

71. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-mediated Diseases (pIMDs)
Description: as for outcome 68
Time Frame: Within 182 days (Days 0-181) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 128 | 64 | 63
Participants | 0 | 0 | 0 | 0

72. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-mediated Diseases (pIMDs)
Description: as for outcome 68
Time Frame: Throughout the entire study period (Day 0 - Day 385)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 128 | 64 | 63
Participants | 0 | 0 | 0 | 0

73. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) - Preliminary Analysis
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Within 21 days (Days 0-20) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 64 | 64 | 63
Participants | 1 | 0 | 0 | 0

74. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) - First Analysis
Description: as for outcome 73
Time Frame: Within 42 days (Days 0-41) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 64 | 64 | 63
Participants | 1 | 0 | 0 | 0

75. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) - Second Analysis
Description: as for outcome 73
Time Frame: Within 42 days (Day 0-41) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 128 | 64 | 63
Participants | 1 | 0 | 0 | 0

76. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 73
Time Frame: Within 182 days (Days 0-181) post vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 128 | 64 | 63
Participants | 1 | 2 | 0 | 0

77. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 73
Time Frame: Throughout the entire study period (Day 0 - Day 385)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
Number analyzed (Participants) | 67 | 128 | 64 | 63
Participants | 2 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 7-day post-vaccination period (Days 0-6). Unsolicited AEs: during the 84-day post-vaccination (Days 0-83). SAEs: during the entire study period (Day 0 - Day 385).
Arm/Group | Arepanrix/F1 Group | Arepanrix/F2 Group | GSK2340273A/F1 Group | GSK2340273A/F2 Group
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/128 | 0/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 2/67 | 2/128 | 0/64 | 0/63
Other Adverse Events (participants affected / at risk) | 61/67 | 125/128 | 54/64 | 55/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arepanrix/F1 Group (N=67) | Arepanrix/F2 Group (N=128) | GSK2340273A/F1 Group (N=64) | GSK2340273A/F2 Group (N=63)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arepanrix/F1 Group (N=67) | Arepanrix/F2 Group (N=128) | GSK2340273A/F1 Group (N=64) | GSK2340273A/F2 Group (N=63)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 11 (12) | 2 (2) | 2 (2)
Chills (General disorders) | 4 (4) | 5 (5) | 2 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 20 (23) | 6 (7) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 27 (36) | 45 (54) | 12 (14) | 11 (14)
Erythema (Skin and subcutaneous tissue disorders) | 14 (18) | 13 (14) | 1 (1) | 2 (2)
Fatigue (General disorders) | 6 (6) | 11 (15) | 4 (7) | 8 (8)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 8 (10) | 3 (4) | 7 (7)
Headache (Nervous system disorders) | 11 (15) | 15 (19) | 4 (4) | 6 (8)
Irritability (Psychiatric disorders) | 28 (41) | 50 (69) | 21 (28) | 17 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (11) | 11 (15) | 3 (4) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (5) | 10 (11) | 4 (6) | 6 (8)
Otitis media (Infections and infestations) | 2 (2) | 8 (10) | 2 (2) | 3 (4)
Pain (General disorders) | 51 (77) | 91 (148) | 34 (50) | 30 (41)
Pyrexia (General disorders) | 32 (36) | 41 (50) | 11 (12) | 10 (11)
Somnolence (Nervous system disorders) | 17 (24) | 42 (51) | 13 (15) | 14 (16)
Swelling (General disorders) | 7 (9) | 15 (17) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 12 (12) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4) | 6 (6) | 2 (2) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.